CLINICAL TRIAL: NCT00548093
Title: A PHASE 2, OPEN-LABEL, TWO ARM TRIAL TO EVALUATE THE EFFICACY OF PF-00299804 IN PATIENTS WITH ADVANCED NSCLC AFTER FAILURE OF AT LEAST ONE PRIOR CHEMOTHERAPY REGIMEN AND FAILURE OF PRIOR TREATMENT WITH ERLOTINIB
Brief Title: PF-00299804 As A Single Agent, In Patients With Advanced Non-Small Cell Lung Cancer Who Have Failed Chemotherapy And Erlotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471002
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: non-small cell lung cancer; advanced; previously treated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): descriptive: adenocarcinoma histology
  Interventions: Drug: PF-00299804
- 2 (Experimental): descriptive: non-adenocarcinoma histology
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — PF-00299804 orally at 45 mg daily, on continuous schedule
  Arms: 1
Drug: PF-00299804 — PF-00299804 orally at 45 mg daily, on continuous schedule
  Arms: 2

SUMMARY:
To assess the antitumor efficacy measured by the objective response rate of oral PF-00299804 taken daily, as single agent in patients with advanced NSCLC who failed at least one chemotherapy + erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small Cell Lung Cancer (NSCLC)
* Prior treatment with and failure of at least one regimen of chemotherapy and erlotinib.
* Prior treatment with no more than two chemotherapy regimens, including adjuvant or combined modality treatment.
* Measurable disease .
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Tissue available for KRAS/ EGFR testing
* Creatinine clearance > 40 cc/min or serum creat < 1.5 x ULN

Exclusion Criteria:

* Chemotherapy
* Radiotherapy
* Biological or investigational agents within 4 weeks of baseline disease assessment.
* Patients who lack of tolerance of erlotinib therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-04-29 (Actual); Primary Completion 2010-03-16 (Actual); Study Completion 2012-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - City of Hope, Duarte, California
  - City of Hope Medical Group, Pasadena, California
  - City of Hope South Pasadena Cancer Center, South Pasadena, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Grady Health Systems, Atlanta, Georgia
  - Emery University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - CCR, National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute/Wayne State University, Detroit, Michigan
  - Lawrence and Idell Weisberg Cancer Treatment Center, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Reckamp KL, Giaccone G, Camidge DR, Gadgeel SM, Khuri FR, Engelman JA, Koczywas M, Rajan A, Campbell AK, Gernhardt D, Ruiz-Garcia A, Letrent S, Liang J, Taylor I, O'Connell JP, Janne PA. A phase 2 trial of dacomitinib (PF-00299804), an oral, irreversible pan-HER (human epidermal growth factor receptor) inhibitor, in patients with advanced non-small cell lung cancer after failure of prior chemotherapy and erlotinib. Cancer. 2014 Apr 15;120(8):1145-54. doi: 10.1002/cncr.28561. Epub 2014 Feb 5. PMID 24501009
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471002&StudyName=PF-00299804%20As%20A%20Single%20Agent%2C%20In%20Patients%20With%20Advanced%20Non-Small%20Cell%20Lung%20Cancer%20%20Who%20Have%20Failed%20Chemotherapy%20And%20Erlotinib

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00299804 (Adenocarcinoma Histology): Participants with adenocarcinoma histology received PF-00299804 tablet 45 milligram (mg) orally once daily in cycles of 21 days until unacceptable toxicity, tumor progression, death, withdrawal from the study or investigator's discretion.
- PF-00299804 (Non-adenocarcinoma Histology): Participants with non-adenocarcinoma histology received PF-00299804 tablet 45 mg orally once daily in cycles of 21 days until unacceptable toxicity, tumor progression, death, withdrawal from the study or investigator's discretion.
Period: Overall Study
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Started | 50 | 16
Completed | 0 | 0
Not Completed | 50 | 16
Not completed — Death | 33 | 13
Not completed — Lost to Follow-up | 3 | 1
Not completed — Objective progression or relapse | 1 | 1
Not completed — Other | 11 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Completed post-treatment follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology) | Total
Number analyzed (Participants) | 50 | 16 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.3) | 65.0 (10.7) | 61.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 2 | 37
  Male | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) in Participants With Adenocarcinoma Histology
Description: BOR:best response recorded from treatment start until disease progression as per Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response: disappearance of all lesions. Partial Response (PR):greater than or equal to (>=)30% decrease in sum of longest diameters (SLDs) of target lesions (TLs) taking as reference baseline SLD. Progressive disease (PD):>=20% increase in SLD of TLs taking as reference smallest SLD since treatment start, or appearance of >=1 new lesion. Stable disease:neither shrinkage for PR nor increase for PD taking as reference smallest SLD since treatment start.
Time Frame: Baseline, end of every even-numbered cycle up to end of treatment (Day 936)
Population: Response-evaluable population included all enrolled participants who received at least 1 dose of study treatment, with adequate baseline tumor assessment and at least 1 on-study tumor assessment after the first dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-00299804 (Adenocarcinoma Histology)
Number analyzed (Participants) | 42
Participants
  Complete response | 0
  Partial response | 2
  Stable or No response | 28
  Objective progression | 12
  Indeterminate | 0

2. Secondary Outcome: Best Overall Response (BOR) in Participants With Non-Adenocarcinoma Histology
Description: BOR: best response recorded from treatment start until disease progression as per RECIST. Complete Response: disappearance of all lesions. PR: >=30% decrease in SLDs of TLs taking as reference baseline SLD. PD: >=20% increase in SLD of TLs taking as reference smallest SLD since treatment start, or appearance of >=1 new lesion. Stable disease: neither shrinkage for PR nor increase for PD taking as reference smallest SLD since treatment start.
Time Frame: Baseline, end of every even-numbered cycle up to end of treatment (Day 936)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 16
Participants
  Complete response | 0
  Partial response | 1
  Stable or no response | 8
  Objective progression | 7
  Indeterminate | 0

3. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline, end of every even-numbered cycle up to end of treatment (Day 936)
Population: DR was calculated for the subgroup of participants from the response-evaluable population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 2 | 1
weeks | 45.2 [24.1 to 66.3] | 12.1 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.

4. Secondary Outcome: Percent Probability of Progression-free Survival (PFS) at Month 6
Description: Probability of being event free (event defined as PD or death due to any cause) at 6 months after the first dose of study treatment. PFS was defined as the time from the first dosing date to the date of first documentation of progression or death due to any cause, whichever occurs first. PFS was calculated as (first event date (if not reached, censored at the last known event-free date) minus first dosing date plus 1). Documentation of progression was determined from objective disease assessment based on RECIST v1.0 criteria. PD was defined as at least a 20% increase in the sum of the longest diameters of the target lesions taking as a reference the smallest sum of the longest diameters recorded since treated started or the appearance of 1 or more new lesions.
Time Frame: Up to 6 months after the start of study medication
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percent chance of being event-free
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 16
percent chance of being event-free | 24.3 [12.4 to 38.4] | 8.0 [0.5 to 29.8]

5. Secondary Outcome: Percent Probability of Overall Survival at Months 6 and 12
Description: Probability of being alive at 6 and 12 months after the first dose of study medication.
Time Frame: Months 6, 12
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percent chance of being alive
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 16
percent chance of being alive
  Month 6 | 71.5 [56.7 to 82.1] | 50.0 [24.5 to 71.0]
  Month 12 | 46.3 [31.4 to 59.9] | 21.9 [5.6 to 44.9]

6. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC (0-24)]
Description: The pharmacokinetic (PK) samples collected between 22-26 hours post dose on Day 1 of Cycle 1 were within the pre-specified time window for the 24-hour post dose sample and were used for calculation of AUC (0-24) on Day 1 of Cycle 1.
Time Frame: 0.5-2, 3-5, 6-8, 22-26 hours post dose on Day 1 of Cycle 1
Population: PK concentration population included all enrolled participants who received at least 1 dose of study treatment and had at least 1 measured plasma concentration. Here, 'N' (overall number of participants analyzed) signifies those participants who were evaluable for the measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 49 | 13
nanogram*hour per milliliter (ng*hr/mL) | 390.8 (165.24) | 397.9 (258.11)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0.5-2, 3-5, 6-8, 22-26 hours post dose on Day 1 of Cycle 1
Population: PK concentration population included all enrolled participants who received at least 1 dose of study treatment and had at least 1 measured plasma concentration. Here, 'N' signifies those participants who were evaluable for the measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 49 | 13
nanogram per milliliter | 22.61 (10.315) | 25.49 (22.533)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0.5-2, 3-5, 6-8, 22-26 hours post dose on Day 1 of Cycle 1
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 49 | 13
hours | 6.08 [3.00 to 25.1] | 6.17 [5.00 to 25.7]

9. Secondary Outcome: Human Epidermal Growth Factor-2 (HER-2) and Epidermal Growth Factor Receptor (EGFR) Levels in Serum
Description: Human epidermal growth factor receptor 2 (HER2) is a transmembrane protein that plays a pivotal role in growth factor signal transduction and epidermal growth factor receptor (EGFR) is a cell surface protein that binds to epidermal growth factor. Levels of the HER-2 and EGFR extracellular domains in serum were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline [pre-dose on Cycle 1 Day 1 (C1D1)], then pre-dose on Day 1 of each cycle, end of treatment (Day 936)
Population: The pharmacodynamic population was defined as members of the ITT (as enrolled) population who had baseline samples submitted per Institutional Review Board (IRB) / Independent Ethics Committee (IEC) approval and participant consent. Here, 'number analyzed' signifies participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 48 | 14
ng/mL
  EGFR: C1D1 | 51.25 (14.86) | 57.28 (15.36)
  EGFR: C2D1: number analyzed (Participants) | 42 | 11
  EGFR: C2D1 | 45.89 (12.42) | 51.05 (11.35)
  EGFR: C3D1: number analyzed (Participants) | 29 | 10
  EGFR: C3D1 | 44.91 (11.43) | 46.79 (7.64)
  EGFR: C4D1: number analyzed (Participants) | 25 | 8
  EGFR: C4D1 | 46.26 (11.7) | 46.72 (9.01)
  EGFR: C5D1: number analyzed (Participants) | 19 | 4
  EGFR: C5D1 | 45.35 (11.32) | 51.2 (9.76)
  EGFR: C6D1: number analyzed (Participants) | 16 | 5
  EGFR: C6D1 | 48.71 (12.01) | 66.52 (20.19)
  EGFR: C7D1: number analyzed (Participants) | 11 | 2
  EGFR: C7D1 | 52.85 (15.6) | 44.29 (9.55)
  EGFR: C8D1: number analyzed (Participants) | 8 | 1
  EGFR: C8D1 | 50.27 (17.05) | 55.93 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EGFR: C9D1: number analyzed (Participants) | 6 | 0
  EGFR: C9D1 | 50.68 (11.41) |
  EGFR: C10D1: number analyzed (Participants) | 6 | 0
  EGFR: C10D1 | 50.45 (11.58) |
  HER2: C1D1 | 9.69 (4.18) | 9.57 (10.27)
  HER2: C2D1: number analyzed (Participants) | 42 | 11
  HER2: C2D1 | 8.2 (3.28) | 9.39 (9.18)
  HER2: C3D1: number analyzed (Participants) | 29 | 10
  HER2: C3D1 | 7.21 (2.31) | 6.46 (2.92)
  HER2: C4D1: number analyzed (Participants) | 25 | 8
  HER2: C4D1 | 7.22 (2.25) | 6.6 (2.44)
  HER2: C5D1: number analyzed (Participants) | 19 | 4
  HER2: C5D1 | 7.02 (1.8) | 8.38 (3.54)
  HER2: C6D1: number analyzed (Participants) | 16 | 5
  HER2: C6D1 | 7.74 (4.55) | 9.9 (7.34)
  HER2: C7D1: number analyzed (Participants) | 11 | 2
  HER2: C7D1 | 6.95 (2.46) | 6.7 (0.42)
  HER2: C8D1: number analyzed (Participants) | 8 | 1
  HER2: C8D1 | 6.61 (2.95) | 11.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  HER2: C9D1: number analyzed (Participants) | 6 | 0
  HER2: C9D1 | 10.23 (11.66) |
  HER2: C10D1: number analyzed (Participants) | 6 | 0
  HER2: C10D1 | 6.00 (2.67) |

10. Secondary Outcome: Number of Participants With Human Epidermal Growth Factor Family (HER-Family) and Kirsten Rat Sarcoma (KRAS) Gene Mutation Status From Free Tumor Deoxy- Ribonucleic Acid (DNA) in Blood at Screening
Description: HER-family is a family of transmembrane protein that plays a pivotal role in growth factor signal transduction and Kirsten Rat Sarcoma (KRAS) gene is an oncogene that encodes a small guanosine triphosphatase (GTPase) transductor protein called KRAS. The mutation status of HER and KRAS genes in tumor DNA present in plasma was determined using a polymerase chain reaction (PCR)-based assay. The gene that is most common in a particular natural population is known as the wild type. Any form of the gene other than the wild type is known as a mutant form. Number of participants with HER-Family and KRAS gene mutation were classified as: wild type, mutant and unknown.
Time Frame: Screening
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 16
Participants
  KRAS mutation: Wild-type | 39 | 15
  KRAS mutation: Mutant | 0 | 0
  KRAS mutation: Unknown | 11 | 1
  HER-2 mutation: Wild-type | 29 | 13
  HER-2 mutation: Mutant | 0 | 0
  HER-2 mutation: Unknown | 21 | 3

11. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ- C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline (C1D1), C2D1 thereafter every subsequent cycle up to C43
Population: As-enrolled population included all participants who were enrolled in the study. Here, 'N' signifies those participants who were evaluable for the measure and 'number analyzed' signifies participants evaluable at each time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 15
units on a scale
  C1D1: GHS | 65.83 (24.99) | 60.56 (25.87)
  C1D1: Physical functioning | 74.70 (22.17) | 70.22 (27.24)
  C1D1: Role functioning | 72.67 (33.46) | 74.44 (32.04)
  C1D1: Emotional Functioning | 77.72 (23.87) | 77.22 (16.51)
  C1D1: Cognitive Functioning | 81.33 (24.89) | 76.67 (28.73)
  C1D1: Social Functioning | 76.33 (30.69) | 67.78 (26.33)
  C1D1: Fatigue | 36.44 (25.99) | 44.44 (26.89)
  C1D1: Nausea, vomiting | 10.33 (18.10) | 10.00 (17.59)
  C1D1: Pain | 30.33 (32.24) | 30.00 (30.99)
  C1D1: Dyspnoea | 30.00 (31.77) | 20.00 (27.60)
  C1D1: Insomnia | 28.00 (31.12) | 35.56 (34.43)
  C1D1: Appetite loss | 22.00 (30.57) | 31.11 (29.46)
  C1D1: Constipation | 16.00 (27.14) | 24.44 (32.04)
  C1D1: Diarrhea | 8.00 (15.88) | 4.44 (11.73)
  C1D1: Financial difficulties: number analyzed (Participants) | 49 | 15
  C1D1: Financial difficulties | 20.41 (32.50) | 22.22 (34.88)
  C2D1: GHS: number analyzed (Participants) | 44 | 13
  C2D1: GHS | 63.83 (24.64) | 63.46 (17.19)
  C2D1: Physical functioning: number analyzed (Participants) | 44 | 13
  C2D1: Physical functioning | 76.82 (22.76) | 79.49 (13.46)
  C2D1: Role functioning: number analyzed (Participants) | 44 | 13
  C2D1: Role functioning | 73.86 (31.00) | 82.05 (27.61)
  C2D1: Emotional Functioning: number analyzed (Participants) | 44 | 13
  C2D1: Emotional Functioning | 79.73 (21.89) | 82.69 (13.38)
  C2D1: Cognitive Functioning: number analyzed (Participants) | 44 | 13
  C2D1: Cognitive Functioning | 81.44 (19.76) | 76.92 (30.08)
  C2D1: Social Functioning: number analyzed (Participants) | 44 | 13
  C2D1: Social Functioning | 79.92 (26.06) | 80.77 (20.24)
  C2D1: Fatigue: number analyzed (Participants) | 44 | 13
  C2D1: Fatigue | 38.51 (27.25) | 41.88 (26.89)
  C2D1: Nausea, vomiting: number analyzed (Participants) | 44 | 13
  C2D1: Nausea, vomiting | 8.71 (12.18) | 6.41 (10.84)
  C2D1: Pain: number analyzed (Participants) | 44 | 13
  C2D1: Pain | 22.35 (25.66) | 20.51 (22.72)
  C2D1: Dyspnoea: number analyzed (Participants) | 44 | 13
  C2D1: Dyspnoea | 20.45 (25.13) | 20.51 (16.88)
  C2D1: Insomnia: number analyzed (Participants) | 44 | 13
  C2D1: Insomnia | 19.70 (28.14) | 17.95 (32.25)
  C2D1: Appetite loss: number analyzed (Participants) | 44 | 13
  C2D1: Appetite loss | 31.82 (34.44) | 38.46 (35.61)
  C2D1: Constipation: number analyzed (Participants) | 44 | 13
  C2D1: Constipation | 12.88 (24.08) | 10.26 (21.01)
  C2D1: Diarrhea: number analyzed (Participants) | 44 | 13
  C2D1: Diarrhea | 54.55 (26.99) | 38.46 (29.96)
  C2D1: Financial difficulties: number analyzed (Participants) | 44 | 13
  C2D1: Financial difficulties | 18.18 (25.37) | 23.08 (34.39)
  C3D1: GHS: number analyzed (Participants) | 40 | 12
  C3D1: GHS | 65.21 (21.84) | 54.86 (25.49)
  C3D1: Physical functioning: number analyzed (Participants) | 39 | 12
  C3D1: Physical functioning | 79.15 (21.59) | 62.22 (30.66)
  C3D1: Role functioning: number analyzed (Participants) | 39 | 12
  C3D1: Role functioning | 73.50 (28.02) | 62.50 (41.51)
  C3D1: Emotional Functioning: number analyzed (Participants) | 40 | 12
  C3D1: Emotional Functioning | 79.17 (23.49) | 71.53 (18.28)
  C3D1: Cognitive Functioning: number analyzed (Participants) | 40 | 12
  C3D1: Cognitive Functioning | 80.83 (24.33) | 73.61 (33.68)
  C3D1: Social Functioning: number analyzed (Participants) | 40 | 12
  C3D1: Social Functioning | 82.92 (21.51) | 65.28 (24.06)
  C3D1: Fatigue: number analyzed (Participants) | 39 | 12
  C3D1: Fatigue | 36.47 (27.92) | 47.22 (28.48)
  C3D1: Nausea, vomiting: number analyzed (Participants) | 39 | 12
  C3D1: Nausea, vomiting | 14.10 (20.43) | 15.28 (15.01)
  C3D1: Pain: number analyzed (Participants) | 40 | 12
  C3D1: Pain | 22.92 (29.40) | 44.44 (35.06)
  C3D1: Dyspnoea: number analyzed (Participants) | 38 | 12
  C3D1: Dyspnoea | 24.56 (32.59) | 22.22 (21.71)
  C3D1: Insomnia: number analyzed (Participants) | 39 | 12
  C3D1: Insomnia | 21.37 (30.09) | 27.78 (39.78)
  C3D1: Appetite loss: number analyzed (Participants) | 39 | 12
  C3D1: Appetite loss | 38.46 (36.30) | 44.44 (38.49)
  C3D1: Constipation: number analyzed (Participants) | 40 | 12
  C3D1: Constipation | 9.17 (21.33) | 25.00 (35.18)
  C3D1: Diarrhea: number analyzed (Participants) | 40 | 12
  C3D1: Diarrhea | 54.17 (28.93) | 38.89 (31.25)
  C3D1: Financial difficulties: number analyzed (Participants) | 39 | 12
  C3D1: Financial difficulties | 17.09 (26.35) | 33.33 (34.82)
  C4D1: GHS: number analyzed (Participants) | 27 | 8
  C4D1: GHS | 69.44 (19.20) | 53.12 (22.69)
  C4D1: Physical functioning: number analyzed (Participants) | 27 | 8
  C4D1: Physical functioning | 82.47 (15.30) | 55.00 (30.81)
  C4D1: Role functioning: number analyzed (Participants) | 27 | 8
  C4D1: Role functioning | 82.10 (23.08) | 56.25 (33.26)
  C4D1: Emotional Functioning: number analyzed (Participants) | 27 | 8
  C4D1: Emotional Functioning | 87.04 (14.86) | 67.71 (24.17)
  C4D1: Cognitive Functioning: number analyzed (Participants) | 27 | 8
  C4D1: Cognitive Functioning | 85.80 (15.12) | 66.67 (30.86)
  C4D1: Social Functioning: number analyzed (Participants) | 27 | 8
  C4D1: Social Functioning | 88.27 (18.95) | 66.67 (26.73)
  C4D1: Fatigue: number analyzed (Participants) | 27 | 8
  C4D1: Fatigue | 30.04 (21.53) | 48.61 (29.66)
  C4D1: Nausea, vomiting: number analyzed (Participants) | 27 | 8
  C4D1: Nausea, vomiting | 5.56 (10.34) | 10.42 (17.68)
  C4D1: Pain: number analyzed (Participants) | 27 | 8
  C4D1: Pain | 17.28 (18.77) | 41.67 (29.55)
  C4D1: Dyspnoea: number analyzed (Participants) | 27 | 8
  C4D1: Dyspnoea | 18.52 (23.27) | 33.33 (35.63)
  C4D1: Insomnia: number analyzed (Participants) | 27 | 8
  C4D1: Insomnia | 13.58 (24.91) | 25.00 (38.83)
  C4D1: Appetite loss: number analyzed (Participants) | 27 | 8
  C4D1: Appetite loss | 29.63 (29.72) | 37.50 (33.03)
  C4D1: Constipation: number analyzed (Participants) | 27 | 8
  C4D1: Constipation | 4.94 (12.07) | 20.83 (35.36)
  C4D1: Diarrhea: number analyzed (Participants) | 27 | 8
  C4D1: Diarrhea | 53.09 (31.02) | 33.33 (25.20)
  C4D1: Financial difficulties: number analyzed (Participants) | 27 | 8
  C4D1: Financial difficulties | 8.64 (19.81) | 25.00 (29.55)
  C5D1: GHS: number analyzed (Participants) | 27 | 7
  C5D1: GHS | 66.67 (22.88) | 54.76 (27.58)
  C5D1: Physical functioning: number analyzed (Participants) | 27 | 7
  C5D1: Physical functioning | 78.52 (18.24) | 63.81 (34.18)
  C5D1: Role functioning: number analyzed (Participants) | 27 | 7
  C5D1: Role functioning | 77.16 (28.17) | 40.48 (40.66)
  C5D1: Emotional Functioning: number analyzed (Participants) | 27 | 7
  C5D1: Emotional Functioning | 80.25 (21.33) | 77.38 (17.82)
  C5D1: Cognitive Functioning: number analyzed (Participants) | 27 | 7
  C5D1: Cognitive Functioning | 83.95 (17.59) | 69.05 (39.00)
  C5D1: Social Functioning: number analyzed (Participants) | 27 | 7
  C5D1: Social Functioning | 81.48 (20.32) | 57.14 (41.79)
  C5D1: Fatigue: number analyzed (Participants) | 27 | 6
  C5D1: Fatigue | 32.51 (24.83) | 53.70 (34.72)
  C5D1: Nausea, vomiting: number analyzed (Participants) | 27 | 7
  C5D1: Nausea, vomiting | 7.41 (14.12) | 9.52 (13.11)
  C5D1: Pain: number analyzed (Participants) | 27 | 7
  C5D1: Pain | 13.58 (21.70) | 50.00 (38.49)
  C5D1: Dyspnoea: number analyzed (Participants) | 27 | 7
  C5D1: Dyspnoea | 25.93 (23.27) | 28.57 (29.99)
  C5D1: Insomnia: number analyzed (Participants) | 27 | 7
  C5D1: Insomnia | 19.75 (26.57) | 33.33 (43.03)
  C5D1: Appetite loss: number analyzed (Participants) | 27 | 7
  C5D1: Appetite loss | 35.80 (31.93) | 33.33 (38.49)
  C5D1: Constipation: number analyzed (Participants) | 27 | 7
  C5D1: Constipation | 7.41 (16.88) | 19.05 (26.23)
  C5D1: Diarrhea: number analyzed (Participants) | 27 | 7
  C5D1: Diarrhea | 46.15 (29.93) | 38.10 (29.99)
  C5D1: Financial difficulties: number analyzed (Participants) | 27 | 7
  C5D1: Financial difficulties | 17.28 (23.33) | 33.33 (38.49)
  C6D1: GHS: number analyzed (Participants) | 18 | 5
  C6D1: GHS | 68.06 (23.44) | 71.67 (11.18)
  C6D1: Physical functioning: number analyzed (Participants) | 18 | 5
  C6D1: Physical functioning | 79.63 (18.50) | 69.33 (36.39)
  C6D1: Role functioning: number analyzed (Participants) | 18 | 5
  C6D1: Role functioning | 80.56 (20.01) | 63.33 (41.50)
  C6D1: Emotional Functioning: number analyzed (Participants) | 18 | 5
  C6D1: Emotional Functioning | 80.09 (20.64) | 81.67 (22.36)
  C6D1: Cognitive Functioning: number analyzed (Participants) | 18 | 5
  C6D1: Cognitive Functioning | 84.26 (17.59) | 83.33 (28.87)
  C6D1: Social Functioning: number analyzed (Participants) | 18 | 5
  C6D1: Social Functioning | 83.33 (19.80) | 83.33 (16.67)
  C6D1: Fatigue: number analyzed (Participants) | 18 | 5
  C6D1: Fatigue | 29.63 (25.57) | 37.78 (20.18)
  C6D1: Nausea, vomiting: number analyzed (Participants) | 18 | 5
  C6D1: Nausea, vomiting | 8.33 (16.42) | 6.67 (14.91)
  C6D1: Pain: number analyzed (Participants) | 18 | 5
  C6D1: Pain | 18.52 (24.85) | 30.00 (27.39)
  C6D1: Dyspnoea: number analyzed (Participants) | 18 | 5
  C6D1: Dyspnoea | 20.37 (25.92) | 13.33 (18.26)
  C6D1: Insomnia: number analyzed (Participants) | 17 | 5
  C6D1: Insomnia | 23.53 (28.30) | 20.00 (18.26)
  C6D1: Appetite loss: number analyzed (Participants) | 18 | 5
  C6D1: Appetite loss | 25.93 (37.15) | 20.00 (44.72)
  C6D1: Constipation: number analyzed (Participants) | 18 | 5
  C6D1: Constipation | 3.70 (10.78) | 26.67 (43.46)
  C6D1: Diarrhea: number analyzed (Participants) | 18 | 5
  C6D1: Diarrhea | 35.19 (21.30) | 20.00 (29.81)
  C6D1: Financial difficulties: number analyzed (Participants) | 18 | 5
  C6D1: Financial difficulties | 11.11 (19.80) | 40.0 (43.46)
  C7D1: GHS: number analyzed (Participants) | 12 | 4
  C7D1: GHS | 65.28 (26.07) | 68.75 (17.18)
  C7D1: Physical functioning: number analyzed (Participants) | 14 | 4
  C7D1: Physical functioning | 79.05 (19.89) | 75.00 (19.15)
  C7D1: Role functioning: number analyzed (Participants) | 14 | 4
  C7D1: Role functioning | 80.95 (25.20) | 70.83 (28.46)
  C7D1: Emotional Functioning: number analyzed (Participants) | 12 | 4
  C7D1: Emotional Functioning | 75.69 (23.15) | 87.50 (15.96)
  C7D1: Cognitive Functioning: number analyzed (Participants) | 12 | 4
  C7D1: Cognitive Functioning | 76.39 (20.67) | 87.50 (25.00)
  C7D1: Social Functioning: number analyzed (Participants) | 12 | 4
  C7D1: Social Functioning | 80.56 (26.43) | 83.33 (19.25)
  C7D1: Fatigue: number analyzed (Participants) | 14 | 4
  C7D1: Fatigue | 34.92 (25.08) | 27.78 (19.25)
  C7D1: Nausea, vomiting: number analyzed (Participants) | 14 | 4
  C7D1: Nausea, vomiting | 5.95 (12.42) | 16.67 (13.61)
  C7D1: Pain: number analyzed (Participants) | 14 | 4
  C7D1: Pain | 14.29 (21.54) | 20.83 (20.97)
  C7D1: Dyspnoea: number analyzed (Participants) | 14 | 4
  C7D1: Dyspnoea | 19.05 (21.54) | 16.67 (19.25)
  C7D1: Insomnia: number analyzed (Participants) | 14 | 4
  C7D1: Insomnia | 26.19 (32.50) | 16.67 (19.25)
  C7D1: Appetite loss: number analyzed (Participants) | 14 | 4
  C7D1: Appetite loss | 23.81 (33.15) | 0.00 (0.00)
  C7D1: Constipation: number analyzed (Participants) | 12 | 4
  C7D1: Constipation | 5.56 (12.97) | 33.33 (27.22)
  C7D1: Diarrhea: number analyzed (Participants) | 12 | 4
  C7D1: Diarrhea | 41.67 (32.18) | 16.67 (19.25)
  C7D1: Financial difficulties: number analyzed (Participants) | 11 | 4
  C7D1: Financial difficulties | 15.15 (22.92) | 33.33 (47.14)
  C8D1: GHS: number analyzed (Participants) | 13 | 3
  C8D1: GHS | 75.00 (19.25) | 61.11 (25.46)
  C8D1: Physical functioning: number analyzed (Participants) | 12 | 3
  C8D1: Physical functioning | 82.22 (13.43) | 57.78 (47.30)
  C8D1: Role functioning: number analyzed (Participants) | 12 | 3
  C8D1: Role functioning | 84.72 (21.86) | 55.56 (50.92)
  C8D1: Emotional Functioning: number analyzed (Participants) | 13 | 3
  C8D1: Emotional Functioning | 80.77 (22.92) | 61.11 (33.68)
  C8D1: Cognitive Functioning: number analyzed (Participants) | 13 | 3
  C8D1: Cognitive Functioning | 75.64 (25.11) | 94.44 (9.62)
  C8D1: Social Functioning: number analyzed (Participants) | 13 | 3
  C8D1: Social Functioning | 87.18 (18.20) | 83.33 (16.67)
  C8D1: Fatigue: number analyzed (Participants) | 12 | 3
  C8D1: Fatigue | 29.63 (24.77) | 55.56 (44.44)
  C8D1: Nausea, vomiting: number analyzed (Participants) | 12 | 3
  C8D1: Nausea, vomiting | 0.00 (0.00) | 16.67 (16.67)
  C8D1: Pain: number analyzed (Participants) | 13 | 3
  C8D1: Pain | 10.26 (14.50) | 33.33 (44.10)
  C8D1: Dyspnoea: number analyzed (Participants) | 12 | 3
  C8D1: Dyspnoea | 22.22 (21.71) | 11.11 (19.25)
  C8D1: Insomnia: number analyzed (Participants) | 12 | 3
  C8D1: Insomnia | 25.00 (35.18) | 11.11 (19.25)
  C8D1: Appetite loss: number analyzed (Participants) | 12 | 3
  C8D1: Appetite loss | 22.22 (32.82) | 33.33 (57.74)
  C8D1: Constipation: number analyzed (Participants) | 12 | 3
  C8D1: Constipation | 8.33 (20.72) | 11.11 (19.25)
  C8D1: Diarrhea: number analyzed (Participants) | 13 | 3
  C8D1: Diarrhea | 33.33 (27.22) | 66.67 (33.33)
  C8D1: Financial difficulties: number analyzed (Participants) | 13 | 3
  C8D1: Financial difficulties | 10.26 (16.01) | 33.33 (57.74)
  C9D1: GHS: number analyzed (Participants) | 9 | 3
  C9D1: GHS | 77.78 (16.14) | 75.00 (14.43)
  C9D1: Physical functioning: number analyzed (Participants) | 9 | 3
  C9D1: Physical functioning | 81.48 (14.44) | 55.56 (50.92)
  C9D1: Role functioning: number analyzed (Participants) | 9 | 3
  C9D1: Role functioning | 88.89 (16.67) | 55.56 (50.92)
  C9D1: Emotional Functioning: number analyzed (Participants) | 9 | 3
  C9D1: Emotional Functioning | 81.48 (22.74) | 61.11 (25.46)
  C9D1: Cognitive Functioning: number analyzed (Participants) | 9 | 3
  C9D1: Cognitive Functioning | 77.78 (27.64) | 100.00 (0.00)
  C9D1: Social Functioning: number analyzed (Participants) | 9 | 3
  C9D1: Social Functioning | 92.59 (12.11) | 72.22 (25.46)
  C9D1: Fatigue: number analyzed (Participants) | 9 | 3
  C9D1: Fatigue | 33.33 (28.33) | 55.56 (50.92)
  C9D1: Nausea, vomiting: number analyzed (Participants) | 9 | 3
  C9D1: Nausea, vomiting | 0.00 (0.00) | 5.56 (9.62)
  C9D1: Pain: number analyzed (Participants) | 9 | 3
  C9D1: Pain | 9.26 (12.11) | 33.33 (57.74)
  C9D1: Dyspnoea: number analyzed (Participants) | 9 | 3
  C9D1: Dyspnoea | 22.22 (23.57) | 22.22 (19.25)
  C9D1: Insomnia: number analyzed (Participants) | 9 | 3
  C9D1: Insomnia | 25.93 (27.78) | 44.44 (50.92)
  C9D1: Appetite loss: number analyzed (Participants) | 9 | 3
  C9D1: Appetite loss | 33.33 (33.33) | 33.33 (57.74)
  C9D1: Constipation: number analyzed (Participants) | 9 | 3
  C9D1: Constipation | 3.70 (11.11) | 11.11 (19.25)
  C9D1: Diarrhea: number analyzed (Participants) | 9 | 3
  C9D1: Diarrhea | 25.93 (22.22) | 33.33 (33.33)
  C9D1: Financial difficulties: number analyzed (Participants) | 9 | 3
  C9D1: Financial difficulties | 7.41 (14.70) | 33.33 (57.74)
  C10D1: GHS: number analyzed (Participants) | 9 | 1
  C10D1: GHS | 74.07 (26.17) | 50.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Physical functioning: number analyzed (Participants) | 9 | 1
  C10D1: Physical functioning | 82.96 (14.57) | 60.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Role functioning: number analyzed (Participants) | 9 | 1
  C10D1: Role functioning | 79.63 (23.24) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Emotional Functioning: number analyzed (Participants) | 9 | 1
  C10D1: Emotional Functioning | 83.33 (20.83) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Cognitive Functioning: number analyzed (Participants) | 9 | 1
  C10D1: Cognitive Functioning | 72.22 (32.27) | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Social Functioning: number analyzed (Participants) | 9 | 1
  C10D1: Social Functioning | 85.19 (19.44) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Fatigue: number analyzed (Participants) | 9 | 1
  C10D1: Fatigue | 35.80 (30.32) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Nausea, vomiting: number analyzed (Participants) | 9 | 1
  C10D1: Nausea, vomiting | 9.26 (27.78) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Pain: number analyzed (Participants) | 9 | 1
  C10D1: Pain | 18.52 (22.74) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Dyspnoea: number analyzed (Participants) | 9 | 1
  C10D1: Dyspnoea | 25.93 (32.39) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Insomnia: number analyzed (Participants) | 9 | 1
  C10D1: Insomnia | 33.33 (33.33) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Appetite loss: number analyzed (Participants) | 9 | 1
  C10D1: Appetite loss | 33.33 (33.33) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Constipation: number analyzed (Participants) | 9 | 1
  C10D1: Constipation | 11.11 (23.57) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Diarrhea: number analyzed (Participants) | 9 | 1
  C10D1: Diarrhea | 37.04 (20.03) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Financial difficulties: number analyzed (Participants) | 9 | 1
  C10D1: Financial difficulties | 11.11 (16.67) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C11D1: GHS: number analyzed (Participants) | 9 | 0
  C11D1: GHS | 72.22 (24.65) |
  C11D1: Physical functioning: number analyzed (Participants) | 9 | 0
  C11D1: Physical functioning | 82.96 (14.95) |
  C11D1: Role functioning: number analyzed (Participants) | 9 | 0
  C11D1: Role functioning | 79.63 (20.03) |
  C11D1: Emotional Functioning: number analyzed (Participants) | 9 | 0
  C11D1: Emotional Functioning | 83.33 (22.44) |
  C11D1: Cognitive Functioning: number analyzed (Participants) | 9 | 0
  C11D1: Cognitive Functioning | 77.78 (25.00) |
  C11D1: Social Functioning: number analyzed (Participants) | 9 | 0
  C11D1: Social Functioning | 90.74 (14.70) |
  C11D1: Fatigue: number analyzed (Participants) | 9 | 0
  C11D1: Fatigue | 24.69 (22.07) |
  C11D1: Nausea, vomiting: number analyzed (Participants) | 9 | 0
  C11D1: Nausea, vomiting | 5.56 (11.79) |
  C11D1: Pain: number analyzed (Participants) | 9 | 0
  C11D1: Pain | 12.96 (18.22) |
  C11D1: Dyspnoea: number analyzed (Participants) | 9 | 0
  C11D1: Dyspnoea | 22.22 (33.33) |
  C11D1: Insomnia: number analyzed (Participants) | 9 | 0
  C11D1: Insomnia | 25.00 (34.50) |
  C11D1: Appetite loss: number analyzed (Participants) | 9 | 0
  C11D1: Appetite loss | 25.93 (32.39) |
  C11D1: Constipation: number analyzed (Participants) | 9 | 0
  C11D1: Constipation | 7.41 (14.70) |
  C11D1: Diarrhea: number analyzed (Participants) | 9 | 0
  C11D1: Diarrhea | 33.33 (16.67) |
  C11D1: Financial difficulties: number analyzed (Participants) | 9 | 0
  C11D1: Financial difficulties | 7.41 (14.70) |
  C12D1: GHS: number analyzed (Participants) | 6 | 0
  C12D1: GHS | 77.78 (27.22) |
  C12D1: Physical functioning: number analyzed (Participants) | 6 | 0
  C12D1: Physical functioning | 85.56 (19.96) |
  C12D1: Role functioning: number analyzed (Participants) | 6 | 0
  C12D1: Role functioning | 91.67 (20.41) |
  C12D1: Emotional Functioning: number analyzed (Participants) | 6 | 0
  C12D1: Emotional Functioning | 81.94 (30.92) |
  C12D1: Cognitive Functioning: number analyzed (Participants) | 6 | 0
  C12D1: Cognitive Functioning | 75.00 (41.83) |
  C12D1: Social Functioning: number analyzed (Participants) | 6 | 0
  C12D1: Social Functioning | 88.89 (20.18) |
  C12D1: Fatigue: number analyzed (Participants) | 6 | 0
  C12D1: Fatigue | 25.93 (37.62) |
  C12D1: Nausea, vomiting: number analyzed (Participants) | 6 | 0
  C12D1: Nausea, vomiting | 5.56 (13.61) |
  C12D1: Pain: number analyzed (Participants) | 6 | 0
  C12D1: Pain | 13.89 (22.15) |
  C12D1: Dyspnoea: number analyzed (Participants) | 6 | 0
  C12D1: Dyspnoea | 27.78 (44.31) |
  C12D1: Insomnia: number analyzed (Participants) | 6 | 0
  C12D1: Insomnia | 33.33 (42.16) |
  C12D1: Appetite loss: number analyzed (Participants) | 6 | 0
  C12D1: Appetite loss | 22.22 (40.37) |
  C12D1: Constipation: number analyzed (Participants) | 6 | 0
  C12D1: Constipation | 0.00 (0.00) |
  C12D1: Diarrhea: number analyzed (Participants) | 6 | 0
  C12D1: Diarrhea | 22.22 (17.21) |
  C12D1: Financial difficulties: number analyzed (Participants) | 6 | 0
  C12D1: Financial difficulties | 5.56 (13.61) |
  C13D1: GHS: number analyzed (Participants) | 3 | 0
  C13D1: GHS | 66.67 (33.33) |
  C13D1: Physical functioning: number analyzed (Participants) | 4 | 0
  C13D1: Physical functioning | 86.67 (12.17) |
  C13D1: Role functioning: number analyzed (Participants) | 4 | 0
  C13D1: Role functioning | 83.33 (33.33) |
  C13D1: Emotional Functioning: number analyzed (Participants) | 3 | 0
  C13D1: Emotional Functioning | 61.11 (33.68) |
  C13D1: Cognitive Functioning: number analyzed (Participants) | 3 | 0
  C13D1: Cognitive Functioning | 55.56 (38.49) |
  C13D1: Social Functioning: number analyzed (Participants) | 3 | 0
  C13D1: Social Functioning | 77.78 (38.49) |
  C13D1: Fatigue: number analyzed (Participants) | 4 | 0
  C13D1: Fatigue | 40.28 (30.56) |
  C13D1: Nausea, vomiting: number analyzed (Participants) | 4 | 0
  C13D1: Nausea, vomiting | 12.50 (25.00) |
  C13D1: Pain: number analyzed (Participants) | 4 | 0
  C13D1: Pain | 25.00 (28.87) |
  C13D1: Dyspnoea: number analyzed (Participants) | 4 | 0
  C13D1: Dyspnoea | 33.33 (38.49) |
  C13D1: Insomnia: number analyzed (Participants) | 4 | 0
  C13D1: Insomnia | 50.00 (43.03) |
  C13D1: Appetite loss: number analyzed (Participants) | 4 | 0
  C13D1: Appetite loss | 41.67 (50.00) |
  C13D1: Constipation: number analyzed (Participants) | 4 | 0
  C13D1: Constipation | 16.67 (19.25) |
  C13D1: Diarrhea: number analyzed (Participants) | 3 | 0
  C13D1: Diarrhea | 11.11 (19.25) |
  C13D1: Financial difficulties: number analyzed (Participants) | 3 | 0
  C13D1: Financial difficulties | 11.11 (19.25) |
  C14D1: GHS: number analyzed (Participants) | 2 | 0
  C14D1: GHS | 79.17 (5.89) |
  C14D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C14D1: Physical functioning | 96.67 (4.71) |
  C14D1: Role functioning: number analyzed (Participants) | 2 | 0
  C14D1: Role functioning | 100.00 (0.00) |
  C14D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C14D1: Emotional Functioning | 100.00 (0.00) |
  C14D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C14D1: Cognitive Functioning | 91.67 (11.79) |
  C14D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C14D1: Social Functioning | 100.00 (0.00) |
  C14D1: Fatigue: number analyzed (Participants) | 2 | 0
  C14D1: Fatigue | 16.67 (7.86) |
  C14D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C14D1: Nausea, vomiting | 8.33 (11.79) |
  C14D1: Pain: number analyzed (Participants) | 2 | 0
  C14D1: Pain | 0.00 (0.00) |
  C14D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C14D1: Dyspnoea | 16.67 (23.57) |
  C14D1: Insomnia: number analyzed (Participants) | 2 | 0
  C14D1: Insomnia | 0.00 (0.00) |
  C14D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C14D1: Appetite loss | 0.00 (0.00) |
  C14D1: Constipation: number analyzed (Participants) | 2 | 0
  C14D1: Constipation | 16.67 (23.57) |
  C14D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C14D1: Diarrhea | 33.33 (0.00) |
  C14D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C14D1: Financial difficulties | 0.00 (0.00) |
  C15D1: GHS: number analyzed (Participants) | 2 | 0
  C15D1: GHS | 91.67 (11.79) |
  C15D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C15D1: Physical functioning | 96.67 (4.71) |
  C15D1: Role functioning: number analyzed (Participants) | 2 | 0
  C15D1: Role functioning | 100.00 (0.00) |
  C15D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C15D1: Emotional Functioning | 95.83 (5.89) |
  C15D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C15D1: Cognitive Functioning | 91.67 (11.79) |
  C15D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C15D1: Social Functioning | 100.00 (0.00) |
  C15D1: Fatigue: number analyzed (Participants) | 2 | 0
  C15D1: Fatigue | 5.56 (7.86) |
  C15D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C15D1: Nausea, vomiting | 0.00 (0.00) |
  C15D1: Pain: number analyzed (Participants) | 2 | 0
  C15D1: Pain | 0.00 (0.00) |
  C15D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C15D1: Dyspnoea | 0.00 (0.00) |
  C15D1: Insomnia: number analyzed (Participants) | 2 | 0
  C15D1: Insomnia | 16.67 (23.57) |
  C15D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C15D1: Appetite loss | 0.00 (0.00) |
  C15D1: Constipation: number analyzed (Participants) | 2 | 0
  C15D1: Constipation | 16.67 (23.57) |
  C15D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C15D1: Diarrhea | 33.33 (0.00) |
  C15D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C15D1: Financial difficulties | 0.00 (0.00) |
  C16D1: GHS: number analyzed (Participants) | 2 | 0
  C16D1: GHS | 87.50 (5.89) |
  C16D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C16D1: Physical functioning | 96.67 (4.71) |
  C16D1: Role functioning: number analyzed (Participants) | 2 | 0
  C16D1: Role functioning | 100.00 (0.00) |
  C16D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C16D1: Emotional Functioning | 87.50 (17.68) |
  C16D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C16D1: Cognitive Functioning | 91.67 (11.79) |
  C16D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C16D1: Social Functioning | 100.00 (0.00) |
  C16D1: Fatigue: number analyzed (Participants) | 2 | 0
  C16D1: Fatigue | 11.11 (15.71) |
  C16D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C16D1: Nausea, vomiting | 0.00 (0.00) |
  C16D1: Pain: number analyzed (Participants) | 2 | 0
  C16D1: Pain | 8.33 (11.79) |
  C16D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C16D1: Dyspnoea | 0.00 (0.00) |
  C16D1: Insomnia: number analyzed (Participants) | 2 | 0
  C16D1: Insomnia | 0.00 (0.00) |
  C16D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C16D1: Appetite loss | 0.00 (0.00) |
  C16D1: Constipation: number analyzed (Participants) | 2 | 0
  C16D1: Constipation | 0.00 (0.00) |
  C16D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C16D1: Diarrhea | 33.33 (0.00) |
  C16D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C16D1: Financial difficulties | 0.00 (0.00) |
  C17D1: GHS: number analyzed (Participants) | 2 | 0
  C17D1: GHS | 87.50 (5.89) |
  C17D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C17D1: Physical functioning | 96.67 (4.71) |
  C17D1: Role functioning: number analyzed (Participants) | 2 | 0
  C17D1: Role functioning | 100.00 (0.00) |
  C17D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C17D1: Emotional Functioning | 87.50 (17.68) |
  C17D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C17D1: Cognitive Functioning | 91.67 (11.79) |
  C17D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C17D1: Social Functioning | 100.00 (0.00) |
  C17D1: Fatigue: number analyzed (Participants) | 2 | 0
  C17D1: Fatigue | 11.11 (15.71) |
  C17D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C17D1: Nausea, vomiting | 8.33 (11.79) |
  C17D1: Pain: number analyzed (Participants) | 2 | 0
  C17D1: Pain | 0.00 (0.00) |
  C17D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C17D1: Dyspnoea | 0.00 (0.00) |
  C17D1: Insomnia: number analyzed (Participants) | 2 | 0
  C17D1: Insomnia | 16.67 (23.57) |
  C17D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C17D1: Appetite loss | 16.67 (23.57) |
  C17D1: Constipation: number analyzed (Participants) | 2 | 0
  C17D1: Constipation | 0.00 (0.00) |
  C17D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C17D1: Diarrhea | 33.33 (0.00) |
  C17D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C17D1: Financial difficulties | 0.00 (0.00) |
  C18D1: GHS: number analyzed (Participants) | 2 | 0
  C18D1: GHS | 79.17 (5.89) |
  C18D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C18D1: Physical functioning | 96.67 (4.71) |
  C18D1: Role functioning: number analyzed (Participants) | 2 | 0
  C18D1: Role functioning | 100.00 (0.00) |
  C18D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C18D1: Emotional Functioning | 87.50 (17.68) |
  C18D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C18D1: Cognitive Functioning | 100.00 (0.00) |
  C18D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C18D1: Social Functioning | 100.00 (0.00) |
  C18D1: Fatigue: number analyzed (Participants) | 2 | 0
  C18D1: Fatigue | 5.56 (7.86) |
  C18D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C18D1: Nausea, vomiting | 8.33 (11.79) |
  C18D1: Pain: number analyzed (Participants) | 2 | 0
  C18D1: Pain | 0.00 (0.00) |
  C18D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C18D1: Dyspnoea | 0.00 (0.00) |
  C18D1: Insomnia: number analyzed (Participants) | 2 | 0
  C18D1: Insomnia | 0.00 (0.00) |
  C18D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C18D1: Appetite loss | 16.67 (23.57) |
  C18D1: Constipation: number analyzed (Participants) | 2 | 0
  C18D1: Constipation | 0.00 (0.00) |
  C18D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C18D1: Diarrhea | 33.33 (0.00) |
  C18D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C18D1: Financial difficulties | 0.00 (0.00) |
  C19D1: GHS: number analyzed (Participants) | 2 | 0
  C19D1: GHS | 87.50 (5.89) |
  C19D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C19D1: Physical functioning | 96.67 (4.71) |
  C19D1: Role functioning: number analyzed (Participants) | 2 | 0
  C19D1: Role functioning | 100.00 (0.00) |
  C19D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C19D1: Emotional Functioning | 95.83 (5.89) |
  C19D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C19D1: Cognitive Functioning | 100.00 (0.00) |
  C19D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C19D1: Social Functioning | 100.00 (0.00) |
  C19D1: Fatigue: number analyzed (Participants) | 2 | 0
  C19D1: Fatigue | 22.22 (0.00) |
  C19D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C19D1: Nausea, vomiting | 0.00 (0.00) |
  C19D1: Pain: number analyzed (Participants) | 2 | 0
  C19D1: Pain | 16.67 (0.00) |
  C19D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C19D1: Dyspnoea | 0.00 (0.00) |
  C19D1: Insomnia: number analyzed (Participants) | 2 | 0
  C19D1: Insomnia | 33.33 (0.00) |
  C19D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C19D1: Appetite loss | 0.00 (0.00) |
  C19D1: Constipation: number analyzed (Participants) | 2 | 0
  C19D1: Constipation | 0.00 (0.00) |
  C19D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C19D1: Diarrhea | 50.00 (23.57) |
  C19D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C19D1: Financial difficulties | 0.00 (0.00) |
  C20D1: GHS: number analyzed (Participants) | 2 | 0
  C20D1: GHS | 83.33 (0.00) |
  C20D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C20D1: Physical functioning | 100.00 (0.00) |
  C20D1: Role functioning: number analyzed (Participants) | 2 | 0
  C20D1: Role functioning | 100.00 (0.00) |
  C20D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C20D1: Emotional Functioning | 100.00 (0.00) |
  C20D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C20D1: Cognitive Functioning | 100.00 (0.00) |
  C20D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C20D1: Social Functioning | 100.00 (0.00) |
  C20D1: Fatigue: number analyzed (Participants) | 2 | 0
  C20D1: Fatigue | 5.56 (7.86) |
  C20D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C20D1: Nausea, vomiting | 0.00 (0.00) |
  C20D1: Pain: number analyzed (Participants) | 2 | 0
  C20D1: Pain | 0.00 (0.00) |
  C20D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C20D1: Dyspnoea | 0.00 (0.00) |
  C20D1: Insomnia: number analyzed (Participants) | 2 | 0
  C20D1: Insomnia | 0.00 (0.00) |
  C20D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C20D1: Appetite loss | 0.00 (0.00) |
  C20D1: Constipation: number analyzed (Participants) | 2 | 0
  C20D1: Constipation | 0.00 (0.00) |
  C20D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C20D1: Diarrhea | 33.33 (0.00) |
  C20D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C20D1: Financial difficulties | 0.00 (0.00) |
  C21D1: GHS: number analyzed (Participants) | 2 | 0
  C21D1: GHS | 83.33 (0.00) |
  C21D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C21D1: Physical functioning | 100.00 (0.00) |
  C21D1: Role functioning: number analyzed (Participants) | 2 | 0
  C21D1: Role functioning | 100.00 (0.00) |
  C21D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C21D1: Emotional Functioning | 91.67 (11.79) |
  C21D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C21D1: Cognitive Functioning | 100.00 (0.00) |
  C21D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C21D1: Social Functioning | 100.00 (0.00) |
  C21D1: Fatigue: number analyzed (Participants) | 2 | 0
  C21D1: Fatigue | 5.56 (7.86) |
  C21D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C21D1: Nausea, vomiting | 0.00 (0.00) |
  C21D1: Pain: number analyzed (Participants) | 2 | 0
  C21D1: Pain | 0.00 (0.00) |
  C21D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C21D1: Dyspnoea | 0.00 (0.00) |
  C21D1: Insomnia: number analyzed (Participants) | 2 | 0
  C21D1: Insomnia | 0.00 (0.00) |
  C21D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C21D1: Appetite loss | 0.00 (0.00) |
  C21D1: Constipation: number analyzed (Participants) | 2 | 0
  C21D1: Constipation | 0.00 (0.00) |
  C21D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C21D1: Diarrhea | 33.33 (0.00) |
  C21D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C21D1: Financial difficulties | 0.00 (0.00) |
  C22D1: GHS: number analyzed (Participants) | 2 | 0
  C22D1: GHS | 83.33 (0.00) |
  C22D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C22D1: Physical functioning | 100.00 (0.00) |
  C22D1: Role functioning: number analyzed (Participants) | 2 | 0
  C22D1: Role functioning | 100.00 (0.00) |
  C22D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C22D1: Emotional Functioning | 91.67 (11.79) |
  C22D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C22D1: Cognitive Functioning | 100.00 (0.00) |
  C22D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C22D1: Social Functioning | 100.00 (0.00) |
  C22D1: Fatigue: number analyzed (Participants) | 2 | 0
  C22D1: Fatigue | 5.56 (7.86) |
  C22D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C22D1: Nausea, vomiting | 0.00 (0.00) |
  C22D1: Pain: number analyzed (Participants) | 2 | 0
  C22D1: Pain | 0.00 (0.00) |
  C22D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C22D1: Dyspnoea | 0.00 (0.00) |
  C22D1: Insomnia: number analyzed (Participants) | 2 | 0
  C22D1: Insomnia | 0.00 (0.00) |
  C22D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C22D1: Appetite loss | 0.00 (0.00) |
  C22D1: Constipation: number analyzed (Participants) | 2 | 0
  C22D1: Constipation | 0.00 (0.00) |
  C22D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C22D1: Diarrhea | 16.67 (23.57) |
  C22D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C22D1: Financial difficulties | 0.00 (0.00) |
  C23D1: GHS: number analyzed (Participants) | 2 | 0
  C23D1: GHS | 83.33 (0.00) |
  C23D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C23D1: Physical functioning | 100.00 (0.00) |
  C23D1: Role functioning: number analyzed (Participants) | 2 | 0
  C23D1: Role functioning | 100.00 (0.00) |
  C23D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C23D1: Emotional Functioning | 87.50 (17.68) |
  C23D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C23D1: Cognitive Functioning | 83.33 (23.57) |
  C23D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C23D1: Social Functioning | 100.00 (0.00) |
  C23D1: Fatigue: number analyzed (Participants) | 2 | 0
  C23D1: Fatigue | 5.56 (7.86) |
  C23D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C23D1: Nausea, vomiting | 0.00 (0.00) |
  C23D1: Pain: number analyzed (Participants) | 2 | 0
  C23D1: Pain | 0.00 (0.00) |
  C23D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C23D1: Dyspnoea | 0.00 (0.00) |
  C23D1: Insomnia: number analyzed (Participants) | 2 | 0
  C23D1: Insomnia | 0.00 (0.00) |
  C23D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C23D1: Appetite loss | 0.00 (0.00) |
  C23D1: Constipation: number analyzed (Participants) | 2 | 0
  C23D1: Constipation | 0.00 (0.00) |
  C23D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C23D1: Diarrhea | 33.33 (0.00) |
  C23D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C23D1: Financial difficulties | 0.00 (0.00) |
  C24D1: GHS: number analyzed (Participants) | 2 | 0
  C24D1: GHS | 83.33 (0.00) |
  C24D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C24D1: Physical functioning | 100.00 (0.00) |
  C24D1: Role functioning: number analyzed (Participants) | 2 | 0
  C24D1: Role functioning | 100.00 (0.00) |
  C24D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C24D1: Emotional Functioning | 83.33 (23.57) |
  C24D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C24D1: Cognitive Functioning | 83.33 (23.57) |
  C24D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C24D1: Social Functioning | 100.00 (0.00) |
  C24D1: Fatigue: number analyzed (Participants) | 2 | 0
  C24D1: Fatigue | 5.56 (7.86) |
  C24D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C24D1: Nausea, vomiting | 8.33 (11.79) |
  C24D1: Pain: number analyzed (Participants) | 2 | 0
  C24D1: Pain | 0.00 (0.00) |
  C24D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C24D1: Dyspnoea | 0.00 (0.00) |
  C24D1: Insomnia: number analyzed (Participants) | 2 | 0
  C24D1: Insomnia | 16.67 (23.57) |
  C24D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C24D1: Appetite loss | 0.00 (0.00) |
  C24D1: Constipation: number analyzed (Participants) | 2 | 0
  C24D1: Constipation | 0.00 (0.00) |
  C24D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C24D1: Diarrhea | 50.00 (23.57) |
  C24D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C24D1: Financial difficulties | 16.67 (23.57) |
  C25D1: GHS: number analyzed (Participants) | 2 | 0
  C25D1: GHS | 83.33 (0.00) |
  C25D1: Physical functioning: number analyzed (Participants) | 2 | 0
  C25D1: Physical functioning | 100.00 (0.00) |
  C25D1: Role functioning: number analyzed (Participants) | 2 | 0
  C25D1: Role functioning | 100.00 (0.00) |
  C25D1: Emotional Functioning: number analyzed (Participants) | 2 | 0
  C25D1: Emotional Functioning | 95.83 (5.89) |
  C25D1: Cognitive Functioning: number analyzed (Participants) | 2 | 0
  C25D1: Cognitive Functioning | 91.67 (11.79) |
  C25D1: Social Functioning: number analyzed (Participants) | 2 | 0
  C25D1: Social Functioning | 100.00 (0.00) |
  C25D1: Fatigue: number analyzed (Participants) | 2 | 0
  C25D1: Fatigue | 11.11 (15.71) |
  C25D1: Nausea, vomiting: number analyzed (Participants) | 2 | 0
  C25D1: Nausea, vomiting | 0.00 (0.00) |
  C25D1: Pain: number analyzed (Participants) | 2 | 0
  C25D1: Pain | 0.00 (0.00) |
  C25D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C25D1: Dyspnoea | 0.00 (0.00) |
  C25D1: Insomnia: number analyzed (Participants) | 2 | 0
  C25D1: Insomnia | 16.67 (23.57) |
  C25D1: Appetite loss: number analyzed (Participants) | 2 | 0
  C25D1: Appetite loss | 16.67 (23.57) |
  C25D1: Constipation: number analyzed (Participants) | 2 | 0
  C25D1: Constipation | 0.00 (0.00) |
  C25D1: Diarrhea: number analyzed (Participants) | 2 | 0
  C25D1: Diarrhea | 50.00 (23.57) |
  C25D1: Financial difficulties: number analyzed (Participants) | 2 | 0
  C25D1: Financial difficulties | 16.67 (23.57) |
  C26D1: GHS: number analyzed (Participants) | 1 | 0
  C26D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C26D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Role functioning: number analyzed (Participants) | 1 | 0
  C26D1: Role functioning | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C26D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C26D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C26D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Fatigue: number analyzed (Participants) | 1 | 0
  C26D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C26D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Pain: number analyzed (Participants) | 1 | 0
  C26D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C26D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Insomnia: number analyzed (Participants) | 1 | 0
  C26D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C26D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Constipation: number analyzed (Participants) | 1 | 0
  C26D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C26D1: Diarrhea | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C26D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: GHS: number analyzed (Participants) | 1 | 0
  C27D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C27D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Role functioning: number analyzed (Participants) | 1 | 0
  C27D1: Role functioning | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C27D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C27D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C27D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Fatigue: number analyzed (Participants) | 1 | 0
  C27D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C27D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Pain: number analyzed (Participants) | 1 | 0
  C27D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C27D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Insomnia: number analyzed (Participants) | 1 | 0
  C27D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C27D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Constipation: number analyzed (Participants) | 1 | 0
  C27D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C27D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C27D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: GHS: number analyzed (Participants) | 1 | 0
  C29D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C29D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Role functioning: number analyzed (Participants) | 1 | 0
  C29D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C29D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C29D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C29D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Fatigue: number analyzed (Participants) | 1 | 0
  C29D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C29D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Pain: number analyzed (Participants) | 1 | 0
  C29D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C29D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Insomnia: number analyzed (Participants) | 1 | 0
  C29D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C29D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Constipation: number analyzed (Participants) | 1 | 0
  C29D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C29D1: Diarrhea | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C29D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: GHS: number analyzed (Participants) | 1 | 0
  C30D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C30D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Role functioning: number analyzed (Participants) | 1 | 0
  C30D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C30D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C30D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C30D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Fatigue: number analyzed (Participants) | 1 | 0
  C30D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C30D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Pain: number analyzed (Participants) | 1 | 0
  C30D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C30D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Insomnia: number analyzed (Participants) | 1 | 0
  C30D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C30D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Constipation: number analyzed (Participants) | 1 | 0
  C30D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C30D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C30D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: GHS: number analyzed (Participants) | 1 | 0
  C31D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C31D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Role functioning: number analyzed (Participants) | 1 | 0
  C31D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C31D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C31D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C31D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Fatigue: number analyzed (Participants) | 1 | 0
  C31D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C31D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Pain: number analyzed (Participants) | 1 | 0
  C31D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C31D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Insomnia: number analyzed (Participants) | 1 | 0
  C31D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C31D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Constipation: number analyzed (Participants) | 1 | 0
  C31D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C31D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C31D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: GHS: number analyzed (Participants) | 1 | 0
  C32D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C32D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Role functioning: number analyzed (Participants) | 1 | 0
  C32D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C32D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C32D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C32D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Fatigue: number analyzed (Participants) | 1 | 0
  C32D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C32D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Pain: number analyzed (Participants) | 1 | 0
  C32D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C32D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Insomnia: number analyzed (Participants) | 1 | 0
  C32D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C32D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Constipation: number analyzed (Participants) | 1 | 0
  C32D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C32D1: Diarrhea | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C32D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: GHS: number analyzed (Participants) | 1 | 0
  C33D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C33D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Role functioning: number analyzed (Participants) | 1 | 0
  C33D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C33D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C33D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C33D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Fatigue: number analyzed (Participants) | 1 | 0
  C33D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C33D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Pain: number analyzed (Participants) | 1 | 0
  C33D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C33D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Insomnia: number analyzed (Participants) | 1 | 0
  C33D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C33D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Constipation: number analyzed (Participants) | 1 | 0
  C33D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C33D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C33D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: GHS: number analyzed (Participants) | 1 | 0
  C34D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C34D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Role functioning: number analyzed (Participants) | 1 | 0
  C34D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C34D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C34D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C34D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Fatigue: number analyzed (Participants) | 1 | 0
  C34D1: Fatigue | 11.11 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C34D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Pain: number analyzed (Participants) | 1 | 0
  C34D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C34D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Insomnia: number analyzed (Participants) | 1 | 0
  C34D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C34D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Constipation: number analyzed (Participants) | 1 | 0
  C34D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C34D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C34D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: GHS: number analyzed (Participants) | 1 | 0
  C35D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C35D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Role functioning: number analyzed (Participants) | 1 | 0
  C35D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C35D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C35D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C35D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Fatigue: number analyzed (Participants) | 1 | 0
  C35D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C35D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Pain: number analyzed (Participants) | 1 | 0
  C35D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C35D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Insomnia: number analyzed (Participants) | 1 | 0
  C35D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C35D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Constipation: number analyzed (Participants) | 1 | 0
  C35D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C35D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C35D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: GHS: number analyzed (Participants) | 1 | 0
  C36D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C36D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Role functioning: number analyzed (Participants) | 1 | 0
  C36D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C36D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C36D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C36D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Fatigue: number analyzed (Participants) | 1 | 0
  C36D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C36D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Pain: number analyzed (Participants) | 1 | 0
  C36D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C36D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Insomnia: number analyzed (Participants) | 1 | 0
  C36D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C36D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Constipation: number analyzed (Participants) | 1 | 0
  C36D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C36D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C36D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: GHS: number analyzed (Participants) | 1 | 0
  C37D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C37D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Role functioning: number analyzed (Participants) | 1 | 0
  C37D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C37D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C37D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C37D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Fatigue: number analyzed (Participants) | 1 | 0
  C37D1: Fatigue | 11.11 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C37D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Pain: number analyzed (Participants) | 1 | 0
  C37D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C37D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Insomnia: number analyzed (Participants) | 1 | 0
  C37D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C37D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Constipation: number analyzed (Participants) | 1 | 0
  C37D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C37D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C37D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: GHS: number analyzed (Participants) | 1 | 0
  C38D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C38D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Role functioning: number analyzed (Participants) | 1 | 0
  C38D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C38D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C38D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C38D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Fatigue: number analyzed (Participants) | 1 | 0
  C38D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C38D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Pain: number analyzed (Participants) | 1 | 0
  C38D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C38D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Insomnia: number analyzed (Participants) | 1 | 0
  C38D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C38D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Constipation: number analyzed (Participants) | 1 | 0
  C38D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C38D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C38D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: GHS: number analyzed (Participants) | 1 | 0
  C39D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C39D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Role functioning: number analyzed (Participants) | 1 | 0
  C39D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C39D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C39D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C39D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Fatigue: number analyzed (Participants) | 1 | 0
  C39D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C39D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Pain: number analyzed (Participants) | 1 | 0
  C39D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C39D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Insomnia: number analyzed (Participants) | 1 | 0
  C39D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C39D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Constipation: number analyzed (Participants) | 1 | 0
  C39D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C39D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C39D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: GHS: number analyzed (Participants) | 1 | 0
  C40D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C40D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Role functioning: number analyzed (Participants) | 1 | 0
  C40D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C40D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C40D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C40D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Fatigue: number analyzed (Participants) | 1 | 0
  C40D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C40D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Pain: number analyzed (Participants) | 1 | 0
  C40D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C40D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Insomnia: number analyzed (Participants) | 1 | 0
  C40D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C40D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Constipation: number analyzed (Participants) | 1 | 0
  C40D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C40D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C40D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: GHS: number analyzed (Participants) | 1 | 0
  C41D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C41D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Role functioning: number analyzed (Participants) | 1 | 0
  C41D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C41D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C41D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C41D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Fatigue: number analyzed (Participants) | 1 | 0
  C41D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C41D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Pain: number analyzed (Participants) | 1 | 0
  C41D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C41D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Insomnia: number analyzed (Participants) | 1 | 0
  C41D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C41D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Constipation: number analyzed (Participants) | 1 | 0
  C41D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C41D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C41D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: GHS: number analyzed (Participants) | 1 | 0
  C42D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C42D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Role functioning: number analyzed (Participants) | 1 | 0
  C42D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C42D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C42D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C42D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Fatigue: number analyzed (Participants) | 1 | 0
  C42D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C42D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Pain: number analyzed (Participants) | 1 | 0
  C42D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C42D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Insomnia: number analyzed (Participants) | 1 | 0
  C42D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C42D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Constipation: number analyzed (Participants) | 1 | 0
  C42D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C42D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C42D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: GHS: number analyzed (Participants) | 1 | 0
  C43D1: GHS | 83.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Physical functioning: number analyzed (Participants) | 1 | 0
  C43D1: Physical functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Role functioning: number analyzed (Participants) | 1 | 0
  C43D1: Role functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Emotional Functioning: number analyzed (Participants) | 1 | 0
  C43D1: Emotional Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Cognitive Functioning: number analyzed (Participants) | 1 | 0
  C43D1: Cognitive Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Social Functioning: number analyzed (Participants) | 1 | 0
  C43D1: Social Functioning | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Fatigue: number analyzed (Participants) | 1 | 0
  C43D1: Fatigue | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Nausea, vomiting: number analyzed (Participants) | 1 | 0
  C43D1: Nausea, vomiting | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Pain: number analyzed (Participants) | 1 | 0
  C43D1: Pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C43D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Insomnia: number analyzed (Participants) | 1 | 0
  C43D1: Insomnia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Appetite loss: number analyzed (Participants) | 1 | 0
  C43D1: Appetite loss | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Constipation: number analyzed (Participants) | 1 | 0
  C43D1: Constipation | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Diarrhea: number analyzed (Participants) | 1 | 0
  C43D1: Diarrhea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Financial difficulties: number analyzed (Participants) | 1 | 0
  C43D1: Financial difficulties | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |

12. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Lung Cancer-13 (QLQ- LC13) Score
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnoea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Baseline (C1D1), C2D1 thereafter every subsequent cycle up to C43
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 15
units on a scale
  C1D1: Dyspnoea: number analyzed (Participants) | 49 | 14
  C1D1: Dyspnoea | 25.85 (22.84) | 26.98 (21.67)
  C1D1: Coughing | 33.33 (30.12) | 33.33 (25.20)
  C1D1: Hemoptysis | 2.00 (10.45) | 4.44 (11.73)
  C1D1: Sore mouth | 3.33 (10.10) | 6.67 (18.69)
  C1D1: Dysphagia | 2.67 (9.13) | 0.00 (0.00)
  C1D1: Peripheral neuropathy | 10.00 (18.13) | 13.33 (24.56)
  C1D1: Alopecia: number analyzed (Participants) | 49 | 15
  C1D1: Alopecia | 8.16 (25.94) | 22.22 (37.09)
  C1D1: Chest pain | 14.67 (27.07) | 20.00 (30.34)
  C1D1: Arm pain | 20.00 (30.12) | 17.78 (33.01)
  C1D1: Other pain | 32.00 (32.96) | 37.78 (33.01)
  C2D1: Dyspnoea: number analyzed (Participants) | 44 | 12
  C2D1: Dyspnoea | 18.69 (20.02) | 26.85 (23.43)
  C2D1: Coughing: number analyzed (Participants) | 44 | 12
  C2D1: Coughing | 19.70 (19.45) | 33.33 (24.62)
  C2D1: Hemoptysis: number analyzed (Participants) | 44 | 12
  C2D1: Hemoptysis | 2.27 (8.50) | 5.56 (12.97)
  C2D1: Sore mouth: number analyzed (Participants) | 44 | 12
  C2D1: Sore mouth | 36.36 (32.00) | 27.78 (23.92)
  C2D1: Dysphagia: number analyzed (Participants) | 44 | 12
  C2D1: Dysphagia | 7.58 (14.13) | 11.11 (16.41)
  C2D1: Peripheral neuropathy: number analyzed (Participants) | 44 | 12
  C2D1: Peripheral neuropathy | 12.12 (20.45) | 13.89 (22.29)
  C2D1: Alopecia: number analyzed (Participants) | 44 | 12
  C2D1: Alopecia | 6.06 (20.68) | 8.33 (15.08)
  C2D1: Chest pain: number analyzed (Participants) | 44 | 12
  C2D1: Chest pain | 10.61 (21.29) | 13.89 (17.16)
  C2D1: Arm pain: number analyzed (Participants) | 44 | 12
  C2D1: Arm pain | 14.39 (20.83) | 19.44 (38.82)
  C2D1: Other pain: number analyzed (Participants) | 44 | 12
  C2D1: Other pain | 22.76 (26.29) | 16.67 (30.15)
  C3D1: Dyspnoea: number analyzed (Participants) | 39 | 12
  C3D1: Dyspnoea | 21.37 (23.69) | 18.52 (14.47)
  C3D1: Coughing: number analyzed (Participants) | 39 | 12
  C3D1: Coughing | 23.08 (20.45) | 41.67 (25.13)
  C3D1: Hemoptysis: number analyzed (Participants) | 40 | 12
  C3D1: Hemoptysis | 1.67 (7.36) | 5.56 (12.97)
  C3D1: Sore mouth: number analyzed (Participants) | 40 | 12
  C3D1: Sore mouth | 30.00 (31.85) | 16.67 (22.47)
  C3D1: Dysphagia: number analyzed (Participants) | 40 | 12
  C3D1: Dysphagia | 11.67 (24.52) | 11.11 (21.71)
  C3D1: Peripheral neuropathy: number analyzed (Participants) | 39 | 12
  C3D1: Peripheral neuropathy | 16.24 (24.03) | 22.22 (25.95)
  C3D1: Alopecia: number analyzed (Participants) | 40 | 12
  C3D1: Alopecia | 4.17 (13.48) | 8.33 (15.08)
  C3D1: Chest pain: number analyzed (Participants) | 40 | 12
  C3D1: Chest pain | 11.67 (23.33) | 19.44 (22.29)
  C3D1: Arm pain: number analyzed (Participants) | 40 | 12
  C3D1: Arm pain | 8.33 (16.45) | 25.00 (32.18)
  C3D1: Other pain: number analyzed (Participants) | 39 | 12
  C3D1: Other pain | 23.08 (26.66) | 33.33 (30.43)
  C4D1: Dyspnoea: number analyzed (Participants) | 26 | 8
  C4D1: Dyspnoea | 15.81 (16.08) | 31.94 (26.85)
  C4D1: Coughing: number analyzed (Participants) | 26 | 8
  C4D1: Coughing | 21.79 (20.96) | 41.67 (23.57)
  C4D1: Hemoptysis: number analyzed (Participants) | 26 | 8
  C4D1: Hemoptysis | 2.56 (9.06) | 4.17 (11.79)
  C4D1: Sore mouth: number analyzed (Participants) | 26 | 8
  C4D1: Sore mouth | 19.23 (19.26) | 20.83 (24.80)
  C4D1: Dysphagia: number analyzed (Participants) | 26 | 8
  C4D1: Dysphagia | 7.69 (14.32) | 16.67 (30.86)
  C4D1: Peripheral neuropathy: number analyzed (Participants) | 26 | 8
  C4D1: Peripheral neuropathy | 19.23 (28.55) | 25.00 (15.43)
  C4D1: Alopecia: number analyzed (Participants) | 26 | 8
  C4D1: Alopecia | 6.41 (21.12) | 4.17 (11.79)
  C4D1: Chest pain: number analyzed (Participants) | 26 | 8
  C4D1: Chest pain | 3.85 (10.86) | 20.83 (30.54)
  C4D1: Arm pain: number analyzed (Participants) | 26 | 8
  C4D1: Arm pain | 7.69 (17.15) | 29.17 (33.03)
  C4D1: Other pain: number analyzed (Participants) | 25 | 8
  C4D1: Other pain | 28.00 (24.87) | 37.50 (27.82)
  C5D1: Dyspnoea: number analyzed (Participants) | 26 | 7
  C5D1: Dyspnoea | 20.51 (17.12) | 20.63 (13.50)
  C5D1: Coughing: number analyzed (Participants) | 26 | 7
  C5D1: Coughing | 25.64 (17.15) | 42.86 (16.27)
  C5D1: Hemoptysis: number analyzed (Participants) | 26 | 7
  C5D1: Hemoptysis | 1.28 (6.54) | 4.76 (12.60)
  C5D1: Sore mouth: number analyzed (Participants) | 26 | 7
  C5D1: Sore mouth | 19.23 (25.25) | 23.81 (25.20)
  C5D1: Dysphagia: number analyzed (Participants) | 26 | 7
  C5D1: Dysphagia | 7.69 (17.15) | 14.29 (26.23)
  C5D1: Peripheral neuropathy: number analyzed (Participants) | 26 | 7
  C5D1: Peripheral neuropathy | 16.67 (27.08) | 19.05 (17.82)
  C5D1: Alopecia: number analyzed (Participants) | 26 | 7
  C5D1: Alopecia | 8.97 (22.23) | 9.52 (16.27)
  C5D1: Chest pain: number analyzed (Participants) | 26 | 7
  C5D1: Chest pain | 8.97 (17.78) | 9.52 (16.27)
  C5D1: Arm pain: number analyzed (Participants) | 26 | 7
  C5D1: Arm pain | 10.26 (22.65) | 23.81 (37.09)
  C5D1: Other pain: number analyzed (Participants) | 25 | 7
  C5D1: Other pain | 21.33 (30.25) | 33.33 (38.49)
  C6D1: Dyspnoea: number analyzed (Participants) | 18 | 5
  C6D1: Dyspnoea | 17.90 (23.84) | 20.00 (14.49)
  C6D1: Coughing: number analyzed (Participants) | 18 | 5
  C6D1: Coughing | 27.78 (20.61) | 20.00 (18.26)
  C6D1: Hemoptysis: number analyzed (Participants) | 18 | 5
  C6D1: Hemoptysis | 3.70 (10.78) | 0.00 (0.00)
  C6D1: Sore mouth: number analyzed (Participants) | 18 | 5
  C6D1: Sore mouth | 22.22 (22.87) | 26.67 (27.89)
  C6D1: Dysphagia: number analyzed (Participants) | 18 | 5
  C6D1: Dysphagia | 3.70 (10.78) | 0.00 (0.00)
  C6D1: Peripheral neuropathy: number analyzed (Participants) | 18 | 5
  C6D1: Peripheral neuropathy | 16.67 (23.57) | 46.67 (38.01)
  C6D1: Alopecia: number analyzed (Participants) | 18 | 5
  C6D1: Alopecia | 11.11 (16.17) | 20.00 (18.26)
  C6D1: Chest pain: number analyzed (Participants) | 18 | 5
  C6D1: Chest pain | 7.41 (18.28) | 0.00 (0.00)
  C6D1: Arm pain: number analyzed (Participants) | 18 | 5
  C6D1: Arm pain | 9.26 (15.36) | 6.67 (14.91)
  C6D1: Other pain: number analyzed (Participants) | 16 | 5
  C6D1: Other pain | 16.67 (24.34) | 40.00 (43.46)
  C7D1: Dyspnoea: number analyzed (Participants) | 14 | 4
  C7D1: Dyspnoea | 17.46 (18.85) | 19.44 (16.67)
  C7D1: Coughing: number analyzed (Participants) | 14 | 4
  C7D1: Coughing | 21.43 (21.11) | 16.67 (19.25)
  C7D1: Hemoptysis: number analyzed (Participants) | 14 | 4
  C7D1: Hemoptysis | 2.38 (8.91) | 0.00 (0.00)
  C7D1: Sore mouth: number analyzed (Participants) | 14 | 4
  C7D1: Sore mouth | 26.19 (26.73) | 16.67 (19.25)
  C7D1: Dysphagia: number analyzed (Participants) | 14 | 4
  C7D1: Dysphagia | 11.90 (21.11) | 8.33 (16.67)
  C7D1: Peripheral neuropathy: number analyzed (Participants) | 14 | 4
  C7D1: Peripheral neuropathy | 19.05 (31.25) | 16.67 (19.25)
  C7D1: Alopecia: number analyzed (Participants) | 14 | 4
  C7D1: Alopecia | 11.90 (16.57) | 8.33 (16.67)
  C7D1: Chest pain: number analyzed (Participants) | 14 | 4
  C7D1: Chest pain | 4.76 (12.10) | 8.33 (16.67)
  C7D1: Arm pain: number analyzed (Participants) | 14 | 4
  C7D1: Arm pain | 11.90 (21.11) | 8.33 (16.67)
  C7D1: Other pain: number analyzed (Participants) | 13 | 4
  C7D1: Other pain | 15.38 (22.01) | 25.00 (31.91)
  C8D1: Dyspnoea: number analyzed (Participants) | 13 | 3
  C8D1: Dyspnoea | 15.38 (14.01) | 29.63 (27.96)
  C8D1: Coughing: number analyzed (Participants) | 13 | 3
  C8D1: Coughing | 28.21 (26.69) | 11.11 (19.25)
  C8D1: Hemoptysis: number analyzed (Participants) | 13 | 3
  C8D1: Hemoptysis | 5.13 (12.52) | 0.00 (0.00)
  C8D1: Sore mouth: number analyzed (Participants) | 13 | 3
  C8D1: Sore mouth | 12.82 (16.88) | 22.22 (19.25)
  C8D1: Dysphagia: number analyzed (Participants) | 13 | 3
  C8D1: Dysphagia | 7.69 (14.62) | 11.11 (19.25)
  C8D1: Peripheral neuropathy: number analyzed (Participants) | 13 | 3
  C8D1: Peripheral neuropathy | 15.38 (22.01) | 33.33 (0.00)
  C8D1: Alopecia: number analyzed (Participants) | 13 | 3
  C8D1: Alopecia | 12.82 (16.88) | 22.22 (19.25)
  C8D1: Chest pain: number analyzed (Participants) | 13 | 3
  C8D1: Chest pain | 7.69 (14.62) | 0.00 (0.00)
  C8D1: Arm pain: number analyzed (Participants) | 12 | 3
  C8D1: Arm pain | 8.33 (15.08) | 11.11 (19.25)
  C8D1: Other pain: number analyzed (Participants) | 13 | 3
  C8D1: Other pain | 23.08 (21.01) | 22.22 (38.49)
  C9D1: Dyspnoea: number analyzed (Participants) | 9 | 3
  C9D1: Dyspnoea | 23.46 (20.37) | 25.93 (23.13)
  C9D1: Coughing: number analyzed (Participants) | 9 | 3
  C9D1: Coughing | 29.63 (20.03) | 11.11 (19.25)
  C9D1: Hemoptysis: number analyzed (Participants) | 9 | 3
  C9D1: Hemoptysis | 3.70 (11.11) | 0.00 (0.00)
  C9D1: Sore mouth: number analyzed (Participants) | 9 | 3
  C9D1: Sore mouth | 7.41 (14.70) | 0.00 (0.00)
  C9D1: Dysphagia: number analyzed (Participants) | 9 | 3
  C9D1: Dysphagia | 11.11 (16.67) | 0.00 (0.00)
  C9D1: Peripheral neuropathy: number analyzed (Participants) | 9 | 3
  C9D1: Peripheral neuropathy | 11.11 (16.67) | 44.44 (19.25)
  C9D1: Alopecia: number analyzed (Participants) | 8 | 3
  C9D1: Alopecia | 8.33 (15.43) | 22.22 (19.25)
  C9D1: Chest pain: number analyzed (Participants) | 9 | 3
  C9D1: Chest pain | 7.41 (14.70) | 0.00 (0.00)
  C9D1: Arm pain: number analyzed (Participants) | 9 | 3
  C9D1: Arm pain | 14.81 (24.22) | 22.22 (38.49)
  C9D1: Other pain: number analyzed (Participants) | 9 | 3
  C9D1: Other pain | 22.22 (23.57) | 55.56 (50.92)
  C10D1: Dyspnoea: number analyzed (Participants) | 9 | 1
  C10D1: Dyspnoea | 23.46 (25.73) | 44.44 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Coughing: number analyzed (Participants) | 9 | 1
  C10D1: Coughing | 25.93 (22.22) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Hemoptysis: number analyzed (Participants) | 9 | 1
  C10D1: Hemoptysis | 3.70 (11.11) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Sore mouth: number analyzed (Participants) | 9 | 1
  C10D1: Sore mouth | 11.11 (23.57) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Dysphagia: number analyzed (Participants) | 9 | 1
  C10D1: Dysphagia | 11.11 (16.67) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Peripheral neuropathy: number analyzed (Participants) | 9 | 1
  C10D1: Peripheral neuropathy | 18.52 (24.22) | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Alopecia: number analyzed (Participants) | 9 | 1
  C10D1: Alopecia | 14.81 (17.57) | 66.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Chest pain: number analyzed (Participants) | 9 | 1
  C10D1: Chest pain | 3.70 (11.11) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Arm pain: number analyzed (Participants) | 9 | 1
  C10D1: Arm pain | 14.81 (24.22) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C10D1: Other pain: number analyzed (Participants) | 9 | 1
  C10D1: Other pain | 22.22 (28.87) | 100.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C11D1: Dyspnoea: number analyzed (Participants) | 9 | 0
  C11D1: Dyspnoea | 23.46 (28.02) |
  C11D1: Coughing: number analyzed (Participants) | 9 | 0
  C11D1: Coughing | 25.93 (22.22) |
  C11D1: Hemoptysis: number analyzed (Participants) | 9 | 0
  C11D1: Hemoptysis | 3.70 (11.11) |
  C11D1: Sore mouth: number analyzed (Participants) | 9 | 0
  C11D1: Sore mouth | 11.11 (23.57) |
  C11D1: Dysphagia: number analyzed (Participants) | 9 | 0
  C11D1: Dysphagia | 0.00 (0.00) |
  C11D1: Peripheral neuropathy: number analyzed (Participants) | 9 | 0
  C11D1: Peripheral neuropathy | 14.81 (33.79) |
  C11D1: Alopecia: number analyzed (Participants) | 9 | 0
  C11D1: Alopecia | 11.11 (16.67) |
  C11D1: Chest pain: number analyzed (Participants) | 9 | 0
  C11D1: Chest pain | 11.11 (16.67) |
  C11D1: Arm pain: number analyzed (Participants) | 9 | 0
  C11D1: Arm pain | 14.81 (24.22) |
  C11D1: Other pain: number analyzed (Participants) | 8 | 0
  C11D1: Other pain | 12.50 (24.80) |
  C12D1: Dyspnoea: number analyzed (Participants) | 6 | 0
  C12D1: Dyspnoea | 22.22 (34.43) |
  C12D1: Coughing: number analyzed (Participants) | 6 | 0
  C12D1: Coughing | 27.78 (25.09) |
  C12D1: Hemoptysis: number analyzed (Participants) | 6 | 0
  C12D1: Hemoptysis | 5.56 (13.61) |
  C12D1: Sore mouth: number analyzed (Participants) | 6 | 0
  C12D1: Sore mouth | 5.56 (13.61) |
  C12D1: Dysphagia: number analyzed (Participants) | 6 | 0
  C12D1: Dysphagia | 0.00 (0.00) |
  C12D1: Peripheral neuropathy: number analyzed (Participants) | 6 | 0
  C12D1: Peripheral neuropathy | 5.56 (13.61) |
  C12D1: Alopecia: number analyzed (Participants) | 6 | 0
  C12D1: Alopecia | 16.67 (18.26) |
  C12D1: Chest pain: number analyzed (Participants) | 6 | 0
  C12D1: Chest pain | 22.22 (34.43) |
  C12D1: Arm pain: number analyzed (Participants) | 6 | 0
  C12D1: Arm pain | 22.22 (34.43) |
  C12D1: Other pain: number analyzed (Participants) | 6 | 0
  C12D1: Other pain | 22.22 (40.37) |
  C13D1: Dyspnoea: number analyzed (Participants) | 4 | 0
  C13D1: Dyspnoea | 27.78 (32.08) |
  C13D1: Coughing: number analyzed (Participants) | 4 | 0
  C13D1: Coughing | 41.67 (16.67) |
  C13D1: Hemoptysis: number analyzed (Participants) | 4 | 0
  C13D1: Hemoptysis | 8.33 (16.67) |
  C13D1: Sore mouth: number analyzed (Participants) | 4 | 0
  C13D1: Sore mouth | 16.67 (19.25) |
  C13D1: Dysphagia: number analyzed (Participants) | 4 | 0
  C13D1: Dysphagia | 8.33 (16.67) |
  C13D1: Peripheral neuropathy: number analyzed (Participants) | 4 | 0
  C13D1: Peripheral neuropathy | 16.67 (33.33) |
  C13D1: Alopecia: number analyzed (Participants) | 4 | 0
  C13D1: Alopecia | 16.67 (19.25) |
  C13D1: Chest pain: number analyzed (Participants) | 4 | 0
  C13D1: Chest pain | 33.33 (38.49) |
  C13D1: Arm pain: number analyzed (Participants) | 4 | 0
  C13D1: Arm pain | 33.33 (38.49) |
  C13D1: Other pain: number analyzed (Participants) | 4 | 0
  C13D1: Other pain | 33.33 (38.46) |
  C14D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C14D1: Dyspnoea | 0.00 (0.00) |
  C14D1: Coughing: number analyzed (Participants) | 2 | 0
  C14D1: Coughing | 33.33 (0.00) |
  C14D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C14D1: Hemoptysis | 0.00 (0.00) |
  C14D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C14D1: Sore mouth | 0.00 (0.00) |
  C14D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C14D1: Dysphagia | 16.67 (23.57) |
  C14D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C14D1: Peripheral neuropathy | 0.00 (0.00) |
  C14D1: Alopecia: number analyzed (Participants) | 2 | 0
  C14D1: Alopecia | 0.00 (0.00) |
  C14D1: Chest pain: number analyzed (Participants) | 2 | 0
  C14D1: Chest pain | 0.00 (0.00) |
  C14D1: Arm pain: number analyzed (Participants) | 2 | 0
  C14D1: Arm pain | 0.00 (0.00) |
  C14D1: Other pain: number analyzed (Participants) | 2 | 0
  C14D1: Other pain | 0.00 (0.00) |
  C15D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C15D1: Dyspnoea | 0.00 (0.00) |
  C15D1: Coughing: number analyzed (Participants) | 2 | 0
  C15D1: Coughing | 33.33 (0.00) |
  C15D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C15D1: Hemoptysis | 0.00 (0.00) |
  C15D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C15D1: Sore mouth | 0.00 (0.00) |
  C15D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C15D1: Dysphagia | 0.00 (0.00) |
  C15D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C15D1: Peripheral neuropathy | 0.00 (0.00) |
  C15D1: Alopecia: number analyzed (Participants) | 2 | 0
  C15D1: Alopecia | 0.00 (0.00) |
  C15D1: Chest pain: number analyzed (Participants) | 2 | 0
  C15D1: Chest pain | 0.00 (0.00) |
  C15D1: Arm pain: number analyzed (Participants) | 2 | 0
  C15D1: Arm pain | 0.00 (0.00) |
  C15D1: Other pain: number analyzed (Participants) | 2 | 0
  C15D1: Other pain | 0.00 (0.00) |
  C16D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C16D1: Dyspnoea | 0.00 (0.00) |
  C16D1: Coughing: number analyzed (Participants) | 2 | 0
  C16D1: Coughing | 16.67 (23.57) |
  C16D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C16D1: Hemoptysis | 0.00 (0.00) |
  C16D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C16D1: Sore mouth | 0.00 (0.00) |
  C16D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C16D1: Dysphagia | 0.00 (0.00) |
  C16D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C16D1: Peripheral neuropathy | 0.00 (0.00) |
  C16D1: Alopecia: number analyzed (Participants) | 2 | 0
  C16D1: Alopecia | 0.00 (0.00) |
  C16D1: Chest pain: number analyzed (Participants) | 2 | 0
  C16D1: Chest pain | 0.00 (0.00) |
  C16D1: Arm pain: number analyzed (Participants) | 2 | 0
  C16D1: Arm pain | 0.00 (0.00) |
  C16D1: Other pain: number analyzed (Participants) | 2 | 0
  C16D1: Other pain | 16.67 (23.57) |
  C17D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C17D1: Dyspnoea | 0.00 (0.00) |
  C17D1: Coughing: number analyzed (Participants) | 2 | 0
  C17D1: Coughing | 33.33 (0.00) |
  C17D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C17D1: Hemoptysis | 0.00 (0.00) |
  C17D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C17D1: Sore mouth | 0.00 (0.00) |
  C17D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C17D1: Dysphagia | 16.67 (23.57) |
  C17D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C17D1: Peripheral neuropathy | 0.00 (0.00) |
  C17D1: Alopecia: number analyzed (Participants) | 2 | 0
  C17D1: Alopecia | 0.00 (0.00) |
  C17D1: Chest pain: number analyzed (Participants) | 2 | 0
  C17D1: Chest pain | 0.00 (0.00) |
  C17D1: Arm pain: number analyzed (Participants) | 2 | 0
  C17D1: Arm pain | 0.00 (0.00) |
  C17D1: Other pain: number analyzed (Participants) | 2 | 0
  C17D1: Other pain | 0.00 (0.00) |
  C18D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C18D1: Dyspnoea | 0.00 (0.00) |
  C18D1: Coughing: number analyzed (Participants) | 2 | 0
  C18D1: Coughing | 50.00 (23.57) |
  C18D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C18D1: Hemoptysis | 0.00 (0.00) |
  C18D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C18D1: Sore mouth | 0.00 (0.00) |
  C18D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C18D1: Dysphagia | 16.67 (23.57) |
  C18D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C18D1: Peripheral neuropathy | 0.00 (0.00) |
  C18D1: Alopecia: number analyzed (Participants) | 2 | 0
  C18D1: Alopecia | 0.00 (0.00) |
  C18D1: Chest pain: number analyzed (Participants) | 2 | 0
  C18D1: Chest pain | 0.00 (0.00) |
  C18D1: Arm pain: number analyzed (Participants) | 2 | 0
  C18D1: Arm pain | 0.00 (0.00) |
  C18D1: Other pain: number analyzed (Participants) | 2 | 0
  C18D1: Other pain | 0.00 (0.00) |
  C19D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C19D1: Dyspnoea | 0.00 (0.00) |
  C19D1: Coughing: number analyzed (Participants) | 2 | 0
  C19D1: Coughing | 33.33 (33.33) |
  C19D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C19D1: Hemoptysis | 0.00 (0.00) |
  C19D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C19D1: Sore mouth | 0.00 (0.00) |
  C19D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C19D1: Dysphagia | 16.67 (23.57) |
  C19D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C19D1: Peripheral neuropathy | 0.00 (0.00) |
  C19D1: Alopecia: number analyzed (Participants) | 2 | 0
  C19D1: Alopecia | 0.00 (0.00) |
  C19D1: Chest pain: number analyzed (Participants) | 2 | 0
  C19D1: Chest pain | 0.00 (0.00) |
  C19D1: Arm pain: number analyzed (Participants) | 2 | 0
  C19D1: Arm pain | 0.00 (0.00) |
  C19D1: Other pain: number analyzed (Participants) | 2 | 0
  C19D1: Other pain | 0.00 (0.00) |
  C20D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C20D1: Dyspnoea | 0.00 (0.00) |
  C20D1: Coughing: number analyzed (Participants) | 2 | 0
  C20D1: Coughing | 33.33 (0.00) |
  C20D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C20D1: Hemoptysis | 0.00 (0.00) |
  C20D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C20D1: Sore mouth | 0.00 (0.00) |
  C20D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C20D1: Dysphagia | 16.67 (23.57) |
  C20D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C20D1: Peripheral neuropathy | 0.00 (0.00) |
  C20D1: Alopecia: number analyzed (Participants) | 2 | 0
  C20D1: Alopecia | 0.00 (0.00) |
  C20D1: Chest pain: number analyzed (Participants) | 2 | 0
  C20D1: Chest pain | 0.00 (0.00) |
  C20D1: Arm pain: number analyzed (Participants) | 2 | 0
  C20D1: Arm pain | 0.00 (0.00) |
  C20D1: Other pain: number analyzed (Participants) | 2 | 0
  C20D1: Other pain | 0.00 (0.00) |
  C21D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C21D1: Dyspnoea | 0.00 (0.00) |
  C21D1: Coughing: number analyzed (Participants) | 2 | 0
  C21D1: Coughing | 33.33 (0.00) |
  C21D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C21D1: Hemoptysis | 0.00 (0.00) |
  C21D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C21D1: Sore mouth | 0.00 (0.00) |
  C21D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C21D1: Dysphagia | 0.00 (0.00) |
  C21D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C21D1: Peripheral neuropathy | 0.00 (0.00) |
  C21D1: Alopecia: number analyzed (Participants) | 2 | 0
  C21D1: Alopecia | 0.00 (0.00) |
  C21D1: Chest pain: number analyzed (Participants) | 2 | 0
  C21D1: Chest pain | 0.00 (0.00) |
  C21D1: Arm pain: number analyzed (Participants) | 2 | 0
  C21D1: Arm pain | 0.00 (0.00) |
  C21D1: Other pain: number analyzed (Participants) | 2 | 0
  C21D1: Other pain | 0.00 (0.00) |
  C22D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C22D1: Dyspnoea | 0.00 (0.00) |
  C22D1: Coughing: number analyzed (Participants) | 2 | 0
  C22D1: Coughing | 33.33 (0.00) |
  C22D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C22D1: Hemoptysis | 0.00 (0.00) |
  C22D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C22D1: Sore mouth | 0.00 (0.00) |
  C22D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C22D1: Dysphagia | 0.00 (0.00) |
  C22D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C22D1: Peripheral neuropathy | 0.00 (0.00) |
  C22D1: Alopecia: number analyzed (Participants) | 2 | 0
  C22D1: Alopecia | 0.00 (0.00) |
  C22D1: Chest pain: number analyzed (Participants) | 2 | 0
  C22D1: Chest pain | 0.00 (0.00) |
  C22D1: Arm pain: number analyzed (Participants) | 2 | 0
  C22D1: Arm pain | 0.00 (0.00) |
  C22D1: Other pain: number analyzed (Participants) | 2 | 0
  C22D1: Other pain | 0.00 (0.00) |
  C23D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C23D1: Dyspnoea | 0.00 (0.00) |
  C23D1: Coughing: number analyzed (Participants) | 2 | 0
  C23D1: Coughing | 33.33 (0.00) |
  C23D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C23D1: Hemoptysis | 0.00 (0.00) |
  C23D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C23D1: Sore mouth | 0.00 (0.00) |
  C23D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C23D1: Dysphagia | 0.00 (0.00) |
  C23D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C23D1: Peripheral neuropathy | 0.00 (0.00) |
  C23D1: Alopecia: number analyzed (Participants) | 2 | 0
  C23D1: Alopecia | 0.00 (0.00) |
  C23D1: Chest pain: number analyzed (Participants) | 2 | 0
  C23D1: Chest pain | 0.00 (0.00) |
  C23D1: Arm pain: number analyzed (Participants) | 2 | 0
  C23D1: Arm pain | 0.00 (0.00) |
  C23D1: Other pain: number analyzed (Participants) | 2 | 0
  C23D1: Other pain | 0.00 (0.00) |
  C24D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C24D1: Dyspnoea | 0.00 (0.00) |
  C24D1: Coughing: number analyzed (Participants) | 2 | 0
  C24D1: Coughing | 33.33 (0.00) |
  C24D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C24D1: Hemoptysis | 0.00 (0.00) |
  C24D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C24D1: Sore mouth | 0.00 (0.00) |
  C24D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C24D1: Dysphagia | 16.67 (23.57) |
  C24D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C24D1: Peripheral neuropathy | 16.67 (23.57) |
  C24D1: Alopecia: number analyzed (Participants) | 2 | 0
  C24D1: Alopecia | 0.00 (0.00) |
  C24D1: Chest pain: number analyzed (Participants) | 2 | 0
  C24D1: Chest pain | 0.00 (0.00) |
  C24D1: Arm pain: number analyzed (Participants) | 2 | 0
  C24D1: Arm pain | 0.00 (0.00) |
  C24D1: Other pain: number analyzed (Participants) | 2 | 0
  C24D1: Other pain | 16.67 (23.57) |
  C25D1: Dyspnoea: number analyzed (Participants) | 2 | 0
  C25D1: Dyspnoea | 0.00 (0.00) |
  C25D1: Coughing: number analyzed (Participants) | 2 | 0
  C25D1: Coughing | 33.33 (0.00) |
  C25D1: Hemoptysis: number analyzed (Participants) | 2 | 0
  C25D1: Hemoptysis | 0.00 (0.00) |
  C25D1: Sore mouth: number analyzed (Participants) | 2 | 0
  C25D1: Sore mouth | 0.00 (0.00) |
  C25D1: Dysphagia: number analyzed (Participants) | 2 | 0
  C25D1: Dysphagia | 16.67 (23.57) |
  C25D1: Peripheral neuropathy: number analyzed (Participants) | 2 | 0
  C25D1: Peripheral neuropathy | 0.00 (0.00) |
  C25D1: Alopecia: number analyzed (Participants) | 2 | 0
  C25D1: Alopecia | 16.67 (23.57) |
  C25D1: Chest pain: number analyzed (Participants) | 2 | 0
  C25D1: Chest pain | 0.00 (0.00) |
  C25D1: Arm pain: number analyzed (Participants) | 2 | 0
  C25D1: Arm pain | 0.00 (0.00) |
  C25D1: Other pain: number analyzed (Participants) | 2 | 0
  C25D1: Other pain | 0.00 (0.00) |
  C26D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C26D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable |
  C26D1: Coughing: number analyzed (Participants) | 1 | 0
  C26D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable |
  C26D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C26D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C26D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C26D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C26D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Alopecia: number analyzed (Participants) | 1 | 0
  C26D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Chest pain: number analyzed (Participants) | 1 | 0
  C26D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Arm pain: number analyzed (Participants) | 1 | 0
  C26D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C26D1: Other pain: number analyzed (Participants) | 1 | 0
  C26D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C27D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Coughing: number analyzed (Participants) | 1 | 0
  C27D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C27D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C27D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C27D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C27D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Alopecia: number analyzed (Participants) | 1 | 0
  C27D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Chest pain: number analyzed (Participants) | 1 | 0
  C27D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Arm pain: number analyzed (Participants) | 1 | 0
  C27D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: Other pain: number analyzed (Participants) | 1 | 0
  C27D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C29D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Coughing: number analyzed (Participants) | 1 | 0
  C29D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C29D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C29D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C29D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C29D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Alopecia: number analyzed (Participants) | 1 | 0
  C29D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Chest pain: number analyzed (Participants) | 1 | 0
  C29D1: Chest pain | 0.00 (0.00) |
  C29D1: Arm pain: number analyzed (Participants) | 1 | 0
  C29D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: Other pain: number analyzed (Participants) | 1 | 0
  C29D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C30D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Coughing: number analyzed (Participants) | 1 | 0
  C30D1: Coughing | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C30D1: Hemoptysis | 0.00 (0.00) |
  C30D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C30D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C30D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C30D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Alopecia: number analyzed (Participants) | 1 | 0
  C30D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Chest pain: number analyzed (Participants) | 1 | 0
  C30D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Arm pain: number analyzed (Participants) | 1 | 0
  C30D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: Other pain: number analyzed (Participants) | 1 | 0
  C30D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C31D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Coughing: number analyzed (Participants) | 1 | 0
  C31D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C31D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C31D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C31D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C31D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Alopecia: number analyzed (Participants) | 1 | 0
  C31D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Chest pain: number analyzed (Participants) | 1 | 0
  C31D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Arm pain: number analyzed (Participants) | 1 | 0
  C31D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: Other pain: number analyzed (Participants) | 1 | 0
  C31D1: Other pain | 0.00 (0.00) |
  C32D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C32D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Coughing: number analyzed (Participants) | 1 | 0
  C32D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C32D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C32D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C32D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C32D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Alopecia: number analyzed (Participants) | 1 | 0
  C32D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Chest pain: number analyzed (Participants) | 1 | 0
  C32D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Arm pain: number analyzed (Participants) | 1 | 0
  C32D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: Other pain: number analyzed (Participants) | 1 | 0
  C32D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C33D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Coughing: number analyzed (Participants) | 1 | 0
  C33D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C33D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C33D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C33D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C33D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Alopecia: number analyzed (Participants) | 1 | 0
  C33D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Chest pain: number analyzed (Participants) | 1 | 0
  C33D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Arm pain: number analyzed (Participants) | 1 | 0
  C33D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: Other pain: number analyzed (Participants) | 1 | 0
  C33D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C34D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Coughing: number analyzed (Participants) | 0 | 0
  C34D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C34D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C34D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C34D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C34D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Alopecia: number analyzed (Participants) | 1 | 0
  C34D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Chest pain: number analyzed (Participants) | 1 | 0
  C34D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Arm pain: number analyzed (Participants) | 1 | 0
  C34D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: Other pain: number analyzed (Participants) | 1 | 0
  C34D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C35D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Coughing: number analyzed (Participants) | 1 | 0
  C35D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C35D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C35D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C35D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C35D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Alopecia: number analyzed (Participants) | 1 | 0
  C35D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Chest pain: number analyzed (Participants) | 1 | 0
  C35D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Arm pain: number analyzed (Participants) | 1 | 0
  C35D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: Other pain: number analyzed (Participants) | 1 | 0
  C35D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable |
  C36D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C36D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Coughing: number analyzed (Participants) | 1 | 0
  C36D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C36D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C36D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C36D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C36D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Alopecia: number analyzed (Participants) | 1 | 0
  C36D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Chest pain: number analyzed (Participants) | 1 | 0
  C36D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Arm pain: number analyzed (Participants) | 1 | 0
  C36D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: Other pain: number analyzed (Participants) | 1 | 0
  C36D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C37D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Coughing: number analyzed (Participants) | 1 | 0
  C37D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C37D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C37D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C37D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C37D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Alopecia: number analyzed (Participants) | 1 | 0
  C37D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Chest pain: number analyzed (Participants) | 1 | 0
  C37D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Arm pain: number analyzed (Participants) | 1 | 0
  C37D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: Other pain: number analyzed (Participants) | 1 | 0
  C37D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C38D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Coughing: number analyzed (Participants) | 1 | 0
  C38D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C38D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C38D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C38D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C38D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Alopecia: number analyzed (Participants) | 1 | 0
  C38D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Chest pain: number analyzed (Participants) | 1 | 0
  C38D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Arm pain: number analyzed (Participants) | 1 | 0
  C38D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: Other pain: number analyzed (Participants) | 1 | 0
  C38D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C39D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Coughing: number analyzed (Participants) | 1 | 0
  C39D1: Coughing | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C39D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C39D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C39D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C39D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Alopecia: number analyzed (Participants) | 1 | 0
  C39D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Chest pain: number analyzed (Participants) | 1 | 0
  C39D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Arm pain: number analyzed (Participants) | 1 | 0
  C39D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: Other pain: number analyzed (Participants) | 1 | 0
  C39D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C40D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Coughing: number analyzed (Participants) | 1 | 0
  C40D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C40D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C40D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C40D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C40D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Alopecia: number analyzed (Participants) | 1 | 0
  C40D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Chest pain: number analyzed (Participants) | 1 | 0
  C40D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Arm pain: number analyzed (Participants) | 1 | 0
  C40D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: Other pain: number analyzed (Participants) | 1 | 0
  C40D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C41D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Coughing: number analyzed (Participants) | 0 | 0
  C41D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C41D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C41D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C41D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C41D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Alopecia: number analyzed (Participants) | 1 | 0
  C41D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Chest pain: number analyzed (Participants) | 1 | 0
  C41D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Arm pain: number analyzed (Participants) | 1 | 0
  C41D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: Other pain: number analyzed (Participants) | 1 | 0
  C41D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C42D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Coughing: number analyzed (Participants) | 1 | 0
  C42D1: Coughing | 33.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C42D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C42D1: Sore mouth | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C42D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C42D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Alopecia: number analyzed (Participants) | 1 | 0
  C42D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Chest pain: number analyzed (Participants) | 1 | 0
  C42D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Arm pain: number analyzed (Participants) | 1 | 0
  C42D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: Other pain: number analyzed (Participants) | 0 | 0
  C43D1: Dyspnoea: number analyzed (Participants) | 1 | 0
  C43D1: Dyspnoea | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Coughing: number analyzed (Participants) | 1 | 0
  C43D1: Coughing | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Hemoptysis: number analyzed (Participants) | 1 | 0
  C43D1: Hemoptysis | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Sore mouth: number analyzed (Participants) | 1 | 0
  C43D1: Sore mouth | 0.00 (0.00) |
  C43D1: Dysphagia: number analyzed (Participants) | 1 | 0
  C43D1: Dysphagia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Peripheral neuropathy: number analyzed (Participants) | 1 | 0
  C43D1: Peripheral neuropathy | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Alopecia: number analyzed (Participants) | 1 | 0
  C43D1: Alopecia | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Chest pain: number analyzed (Participants) | 1 | 0
  C43D1: Chest pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Arm pain: number analyzed (Participants) | 1 | 0
  C43D1: Arm pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: Other pain: number analyzed (Participants) | 1 | 0
  C43D1: Other pain | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |

13. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: Self-administered questionnaire to measure health-related quality of life (QoL) of adult participants suffering from skin disease; 10 questions concerning participants' perception of impact of their disease over last week encompassing aspects such as symptoms or feelings, daily activities, leisure, work or school, personal relationships and treatment. Questions scored on a 4-point Likert scale: 0 (not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual questions (0-3) were added to yield a total score (0-30); higher score = greater impairment of participant's QoL.
Time Frame: Baseline (C1D1), C2D1 thereafter every subsequent cycle up to C43
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 15
units on a scale
  C1D1 | 0.38 (0.54) | 0.80 (1.52)
  C2D1: number analyzed (Participants) | 44 | 13
  C2D1 | 3.34 (4.37) | 2.08 (2.22)
  C3D1: number analyzed (Participants) | 40 | 12
  C3D1 | 4.08 (4.31) | 3.08 (3.99)
  C4D1: number analyzed (Participants) | 27 | 8
  C4D1 | 3.56 (3.62) | 5.13 (5.06)
  C5D1: number analyzed (Participants) | 27 | 7
  C5D1 | 4.67 (4.12) | 6.00 (7.62)
  C6D1: number analyzed (Participants) | 18 | 5
  C6D1 | 4.39 (4.65) | 6.00 (6.40)
  C7D1: number analyzed (Participants) | 14 | 4
  C7D1 | 4.00 (5.28) | 5.00 (6.06)
  C8D1: number analyzed (Participants) | 13 | 3
  C8D1 | 3.31 (3.57) | 3.67 (3.21)
  C9D1: number analyzed (Participants) | 9 | 2
  C9D1 | 1.78 (2.49) | 2.50 (3.54)
  C10D1: number analyzed (Participants) | 9 | 1
  C10D1 | 2.22 (2.54) | 8.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  C11D1: number analyzed (Participants) | 9 | 0
  C11D1 | 2.78 (3.35) |
  C12D1: number analyzed (Participants) | 6 | 0
  C12D1 | 2.00 (3.95) |
  C13D1: number analyzed (Participants) | 4 | 0
  C13D1 | 4.00 (3.65) |
  C14D1: number analyzed (Participants) | 2 | 0
  C14D1 | 1.50 (0.71) |
  C15D1: number analyzed (Participants) | 2 | 0
  C15D1 | 1.00 (1.41) |
  C16D1: number analyzed (Participants) | 2 | 0
  C16D1 | 2.00 (0.00) |
  C17D1: number analyzed (Participants) | 2 | 0
  C17D1 | 0.50 (0.71) |
  C18D1: number analyzed (Participants) | 2 | 0
  C18D1 | 0.50 (0.71) |
  C19D1: number analyzed (Participants) | 2 | 0
  C19D1 | 1.00 (1.41) |
  C20D1: number analyzed (Participants) | 2 | 0
  C20D1 | 0.50 (0.71) |
  C21D1: number analyzed (Participants) | 2 | 0
  C21D1 | 1.00 (1.41) |
  C22D1: number analyzed (Participants) | 2 | 0
  C22D1 | 1.00 (1.41) |
  C23D1: number analyzed (Participants) | 2 | 0
  C23D1 | 8.00 (11.31) |
  C24D1: number analyzed (Participants) | 2 | 0
  C24D1 | 1.00 (1.41) |
  C25D1: number analyzed (Participants) | 2 | 0
  C25D1 | 3.00 (0.00) |
  C26D1: number analyzed (Participants) | 1 | 0
  C26D1 | 2.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C27D1: number analyzed (Participants) | 1 | 0
  C27D1 | 1.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C29D1: number analyzed (Participants) | 1 | 0
  C29D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C30D1: number analyzed (Participants) | 1 | 0
  C30D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C31D1: number analyzed (Participants) | 1 | 0
  C31D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C32D1: number analyzed (Participants) | 1 | 0
  C32D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C33D1: number analyzed (Participants) | 1 | 0
  C33D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C34D1: number analyzed (Participants) | 1 | 0
  C34D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C35D1: number analyzed (Participants) | 1 | 0
  C35D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C36D1: number analyzed (Participants) | 1 | 0
  C36D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C37D1: number analyzed (Participants) | 1 | 0
  C37D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C38D1: number analyzed (Participants) | 1 | 0
  C38D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C39D1: number analyzed (Participants) | 1 | 0
  C39D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C40D1: number analyzed (Participants) | 1 | 0
  C40D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C41D1: number analyzed (Participants) | 1 | 0
  C41D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C42D1: number analyzed (Participants) | 1 | 0
  C42D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  C43D1: number analyzed (Participants) | 1 | 0
  C43D1 | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. |

14. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: PFS is defined as time in weeks from randomization to the first documentation of objective tumor progression or death due to any cause. PFS was calculated as = (first event date minus randomization date plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Month 6
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PF-00299804 (Adenocarcinoma Histology): Participants with adenocarcinoma histology received PF-00299804 tablet 45 milligram (mg) orally once daily in cycles of 21 days up to 1 year or until unacceptable toxicity, tumor progression, death or investigator's discretion.
- PF-00299804 (Non-adenocarcinoma Histology): Participants with non-adenocarcinoma histology received PF-00299804 tablet 45 mg orally once daily in cycles of 21 days up to 1 year or until unacceptable toxicity, tumor progression, death or investigator's discretion.
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Number analyzed (Participants) | 50 | 16
percentage of participants | 24.3 [12.4 to 38.4] | 8.0 [0.5 to 29.8]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00299804 (Adenocarcinoma Histology) | PF-00299804 (Non-adenocarcinoma Histology)
Serious Adverse Events (participants affected / at risk) | 9/50 | 6/16
Other Adverse Events (participants affected / at risk) | 50/50 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 (Adenocarcinoma Histology) (N=50) | PF-00299804 (Non-adenocarcinoma Histology) (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 3 | 0
Cystitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 (Adenocarcinoma Histology) (N=50) | PF-00299804 (Non-adenocarcinoma Histology) (N=16)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Blepharitis (Eye disorders) | 2 | 1
Conjunctivitis (Eye disorders) | 3 | 1
Dry eye (Eye disorders) | 1 | 2
Eye discharge (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Atrophic glossitis (Gastrointestinal disorders) | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 44 | 13
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 6
Oral pain (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 13 | 3
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 1
Tongue dry (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 3
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 4 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 31 | 7
Gait disturbance (General disorders) | 1 | 1
Injection site pain (General disorders) | 1 | 0
Mass (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 4 | 3
Mucous membrane disorder (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 4 | 2
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 2 | 1
Localised infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 5 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time (Investigations) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 1
Blood bicarbonate (Investigations) | 1 | 0
Blood creatinine (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 2 | 1
International normalised ratio (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 7 | 3
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Reading disorder (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 3 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 33 | 12
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 7
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 12 | 4
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 6 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Results for PK parameters to be assessed using nonlinear mixed effects modelling (NONMEM) are not provided because of change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.